

A PHASE 3, RANDOMIZED, DOUBLE-BLIND, PLACEBO-CONTROLLED STUDY TO EVALUATE THE SAFETY, TOLERABILITY, AND IMMUNOGENICITY OF RESPIRATORY SYNCYTIAL VIRUS PREFUSION F SUBUNIT VACCINE WHEN COADMINISTERED WITH SEASONAL INACTIVATED INFLUENZA VACCINE IN ADULTS ≥65 YEARS OF AGE

**Study Intervention Number:** PF-06928316

**Study Intervention Name:** Respiratory Syncytial Virus (RSV) Vaccine

**US IND Number:** 017931

**EudraCT Number:** N/A

ClinicalTrials.gov ID: NCT05301322

**Protocol Number:** C3671006

Phase: 3

**Brief Title:** Safety and Immunogenicity of RSVpreF Coadministered With SIIV in Adults ≥65 Years of Age

This document and accompanying materials contain confidential information belonging to Pfizer. Except as otherwise agreed to in writing, by accepting or reviewing these documents, you agree to hold this information in confidence and not copy or disclose it to others (except where required by applicable law) or use it for unauthorized purposes. In the event of any actual or suspected breach of this obligation, Pfizer must be promptly notified.

# **Document History**

| Document | Version Date |
|----------------------|----------------|
| Original protocol | 30 August 2021 |
| Protocol amendment 1 | 29 August 2022 |

This amendment incorporates all revisions to date, including amendments made at the request of country health authorities and IRBs/ECs and any protocol administrative change letter(s).

## **Protocol Amendment Summary of Changes Table**

# Amendment 1 (29 August 2022)

**Overall Rationale for the Amendment:** Sample size was modified because of operational delays impacting the potential pool of eligible participants.

| Section # and Name | Description of Change | Brief Rationale | Substantial or<br>Nonsubstantial |
|---|---|---|---|
| Section 1.1 Synopsis Section 1.2 Study Design Schema Section 4.1 Overall Design | Number of participants changed from 2230 to 1400 and group size from 1115 to 700 | Change in sample size | Substantial |
| Table 6 Primary Endpoint<br>Analysis | Modified the statement for declaring immunogenicity equivalence statement | Change in sample size | Substantial |
| Sections 9.1.2.1, 9.1.2.2<br>Statistical Hypotheses | Modified statistical hypothesis for RSV and SIIV immunogenicity | Change in sample size | Substantial |
| Section 9.5 Sample Size<br>Determination | Provided the rationale for changing the sample size and modified the power calculation | Change in sample size | Substantial |
| Table 9 Sample Size<br>Determination | Adjusted the power for noninferiority | Change in sample size | Substantial |
| Title Page | Added clinical trial number | Missing information | Nonsubstantial |
| Document History | Added Amendment 1 | Tracking document history | Nonsubstantial |
| Summary of Changes Table | New | Lists the changes incorporated into Amendment 1 | Nonsubstantial |
| Section 2.2.1 Clinical<br>Overview | Updated RSV program study details | To include the latest data | Nonsubstantial |

| Section # and Name | Description of Change | Brief Rationale | Substantial or<br>Nonsubstantial |
|---|---|---|---|
| Section 6.10.3 Permitted<br>Nonstudy Vaccines and<br>Medications | Clarified permitted use of corticosteroids | Incorporation of PACL 1 | Nonsubstantial |
| Section 6.10.4 Recording<br>Nonstudy Vaccinations and<br>Concomitant Medications | Combined the 2 statements on<br>COVID-19 vaccination record<br>keeping into a single statement for<br>clarification purposes only | Incorporation of PACL 1 | Nonsubstantial |
| Section 10.1.3 Informed<br>Consent Process | Clarified text regarding the need to reconsent participants | Protocol template change | Nonsubstantial |
| Appendix 8 Abbreviations | Changed msLRTI to LRTI<br>Added GMC | Reflects change to<br>term as done in Study<br>C3671013, added<br>missing entry | Nonsubstantial |
| Throughout document | Formatting modifications | Style change | Nonsubstantial |
| Section 9 Statistical<br>Considerations, Table 5 to<br>Table 9 | Removed abbreviations from footnote | Style change | Nonsubstantial |

# **TABLE OF CONTENTS**

| LIST OF TABLES | 9 |
|---|---|
| 1. PROTOCOL SUMMARY | 10 |
| 1.1. Synopsis | 10 |
| 1.2. Study Design Schema. | 14 |
| 1.3. Schedule of Activities | 15 |
| 2. INTRODUCTION | 16 |
| 2.1. Study Rationale | 17 |
| 2.2. Background | 17 |
| 2.2.1. Clinical Overview | 17 |
| 2.3. Benefit/Risk Assessment. | 19 |
| 2.3.1. Risk Assessment | 20 |
| 2.3.2. Benefit Assessment | 22 |
| 2.3.3. Overall Benefit/Risk Conclusion | 22 |
| 3. OBJECTIVES, ENDPOINTS, AND ESTIMANDS | 22 |
| 4. STUDY DESIGN | 24 |
| 4.1. Overall Design | 24 |
| 4.2. Scientific Rationale for Study Design | 25 |
| 4.2.1. Choice of Contraception/Barrier Requirements | 25 |
| 4.3. Justification for Dose | 25 |
| 4.4. End of Study Definition | 26 |
| 5. STUDY POPULATION | 26 |
| 5.1. Inclusion Criteria | 26 |
| 5.2. Exclusion Criteria. | 27 |
| 5.3. Lifestyle Considerations | 29 |
| 5.3.1. Contraception | 29 |
| 5.4. Screen Failures | 29 |
| 5.5. Criteria for Temporarily Delaying Enrollment/Randomization/Administration of Study Intervention | 29 |
| 6. STUDY INTERVENTION(S) AND CONCOMITANT THERAPY | 30 |
| 6.1. Study Intervention(s) Administered | 30 |
| 6.1.1. Respiratory Syncytial Virus Stabilized Prefusion F Subunit Vaccine | 30 |

| 6.1.2. Concomitant Seasonal Inactivated Influenza Vaccine | 31 |
|---|---|
| 6.2. Administration | 31 |
| 6.3. Medical Devices | 32 |
| 6.4. Preparation, Handling, Storage, and Accountability | 32 |
| 6.4.1. Preparation and Dispensing | 33 |
| 6.5. Measures to Minimize Bias: Randomization and Blinding | 33 |
| 6.5.1. Randomization to Study Intervention | 33 |
| 6.5.2. Blinding Arrangements | 34 |
| 6.5.2.1. Blinding of Study Site Personnel | 34 |
| 6.5.2.2. Blinding of the Sponsor | 34 |
| 6.5.3. Breaking the Blind | 34 |
| 6.6. Study Intervention Compliance | 34 |
| 6.7. Dose Modification. | 34 |
| 6.8. Continued Access to Study Intervention After the End of the Study | 35 |
| 6.9. Treatment of Overdose | 35 |
| 6.10. Concomitant Therapy | 35 |
| 6.10.1. Prohibited Concomitant Vaccinations and Medications | 35 |
| 6.10.2. Withholding Periods for Concomitant Vaccinations and Medications | 35 |
| 6.10.3. Permitted Nonstudy Vaccines and Medications During the Study | 36 |
| 6.10.4. Recording Nonstudy Vaccinations and Concomitant Medications | 36 |
| 7. DISCONTINUATION OF STUDY INTERVENTION AND PARTICIPANT DISCONTINUATION/WITHDRAWAL | 37 |
| 7.1. Discontinuation of Study Intervention | 37 |
| 7.2. Participant Discontinuation/Withdrawal From the Study | 37 |
| 7.2.1. Withdrawal of Consent | 38 |
| 7.3. Lost to Follow-Up | 38 |
| 8. STUDY ASSESSMENTS AND PROCEDURES | 39 |
| 8.1. Efficacy and/or Immunogenicity Assessments | 39 |
| 8.1.1. Efficacy Assessments | 39 |
| 8.1.2. Immunogenicity Assessments | 40 |
| 8.1.2.1. Blood Collection | 40 |

| 8.1.2.2. RSV Vaccine Antibody Testing | 40 |
|---|---|
| 8.1.2.3. SIIV Immune Response Testing | 40 |
| 8.1.2.4. Exploratory Assays, Including Immunogenicity Assessments and Assay Development | 40 |
| 8.1.3. Biological Samples | 41 |
| 8.2. Safety Assessments | 41 |
| 8.2.1. Physical Examinations | 41 |
| 8.2.2. Vital Signs | 41 |
| 8.2.3. Electronic Diary | 41 |
| 8.2.3.1. Local Reactions – Reactogenicity | 42 |
| 8.2.3.2. Systemic Events | 43 |
| 8.2.3.3. Fever Monitoring | 45 |
| 8.2.4. Clinical Safety Laboratory Assessments | 45 |
| 8.2.5. Pregnancy Testing | 45 |
| 8.3. Adverse Events, Serious Adverse Events, and Other Safety Reporting | 45 |
| 8.3.1. Time Period and Frequency for Collecting AE and SAE Information | 46 |
| 8.3.1.1. Reporting SAEs to Pfizer Safety | 47 |
| 8.3.1.2. Recording Nonserious AEs and SAEs on the CRF | 47 |
| 8.3.2. Method of Detecting AEs and SAEs | 47 |
| 8.3.3. Follow-Up of AEs and SAEs | 47 |
| 8.3.4. Regulatory Reporting Requirements for SAEs | 47 |
| 8.3.5. Environmental Exposure, Exposure During Pregnancy or Breastfeeding, and Occupational Exposure | 48 |
| 8.3.5.1. Exposure During Pregnancy | 48 |
| 8.3.5.2. Exposure During Breastfeeding | 50 |
| 8.3.5.3. Occupational Exposure | 50 |
| 8.3.6. Cardiovascular and Death Events | 50 |
| 8.3.7. Disease-Related Events and/or Disease-Related Outcomes Not Qualifying as AEs or SAEs | 50 |
| 8.3.8. Adverse Events of Special Interest | 50 |
| 8.3.9. Medical Device Deficiencies | 51 |
| 8.3.9.1. Time Period for Detecting Medical Device Deficiencies | 51 |

| 8.3.9.2. Follow-Up of Medical Device Deficiencies | 51 |
|---|---|
| 8.3.9.3. Prompt Reporting of Device Deficiencies to the Sponsor | 51 |
| 8.3.9.4. Regulatory Reporting Requirements for Device Deficiencies | 52 |
| 8.3.10. Medication Errors | 52 |
| 8.4. Pharmacokinetics | 53 |
| 8.5. Genetics | 53 |
| 8.6. Biomarkers | 53 |
| 8.7. Immunogenicity Assessments | 53 |
| 8.8. Health Economics | 53 |
| 8.9. Study Procedures | 54 |
| 8.9.1. Visit 1 – Vaccination 1 (Clinic, Day 1) | 54 |
| 8.9.2. Visit 2 – Vaccination 2 (Clinic, 28 to 35 Days After Visit 1) | 56 |
| 8.9.3. Visit 3 Follow-Up After Vaccination 2 (Clinic, 28 to 35 Days After Visit 2) | 57 |
| 8.9.4. Unscheduled Reactogenicity Visits for a Grade 3 or Suspected Grade 4 Reaction. | 58 |
| 9. STATISTICAL CONSIDERATIONS | 59 |
| 9.1. Statistical Hypotheses | 59 |
| 9.1.1. Estimands | 59 |
| 9.1.2. Statistical Hypotheses | 60 |
| 9.1.2.1. Statistical Hypothesis for Primary RSV Immunogenicity | 60 |
| 9.1.2.2. Statistical Hypothesis for SIIV Immunogenicity | 60 |
| 9.1.3. Multiplicity Adjustment | 60 |
| 9.2. Analysis Sets | 61 |
| 9.3. Statistical Analyses | 61 |
| 9.3.1. General Considerations | 61 |
| 9.3.1.1. Analyses for Binary Data | 62 |
| 9.3.1.2. Analyses for Continuous Data | 62 |
| 9.3.2. Primary Endpoint(s) | 63 |
| 9.3.3. Secondary Endpoint(s) | 64 |
| 9.3.4. Exploratory Endpoint(s) | 64 |

| 9.4. Interim Analyses | 64 |
|---|---|
| 9.5. Sample Size Determination | 64 |
| 10. SUPPORTING DOCUMENTATION AND OPERATIONAL CONSIDERATIONS | 66 |
| 10.1. Appendix 1: Regulatory, Ethical, and Study Oversight Considerations | 66 |
| 10.1.1. Regulatory and Ethical Considerations | 66 |
| 10.1.1.1. Reporting of Safety Issues and Serious Breaches of the Protocol or ICH GCP | 66 |
| 10.1.2. Financial Disclosure | 67 |
| 10.1.3. Informed Consent Process | 67 |
| 10.1.4. Data Protection | 68 |
| 10.1.5. Committees Structure | 68 |
| 10.1.5.1. Data Monitoring Committee | 68 |
| 10.1.6. Dissemination of Clinical Study Data | 68 |
| 10.1.7. Data Quality Assurance | 70 |
| 10.1.8. Source Documents | 71 |
| 10.1.9. Study and Site Start and Closure | 71 |
| 10.1.10. Publication Policy | 72 |
| 10.1.11. Sponsor's Qualified Medical Personnel | 73 |
| 10.2. Appendix 2: Adverse Events: Definitions and Procedures for Recording, Evaluating, Follow-Up, and Reporting | 74 |
| 10.2.1. Definition of AE | 74 |
| 10.2.2. Definition of an SAE | 75 |
| 10.2.3. Recording/Reporting and Follow-Up of AEs and/or SAEs During the Active Collection Period | 77 |
| 10.2.4. Reporting of SAEs | 80 |
| 10.3. Appendix 3: Contraceptive and Barrier Guidance | 81 |
| 10.3.1. Male Participant Reproductive Inclusion Criteria | 81 |
| 10.3.2. Female Participant Reproductive Inclusion Criteria | 81 |
| 10.3.3. Woman of Childbearing Potential | 81 |
| 10.3.4. Contraception Methods | 82 |
| 10.4. Appendix 4: Liver Safety: Suggested Actions and Follow-Up Assessments . | 83 |

| Defi | ppendix 5: AEs, ADEs, SAEs, SADEs, USADEs, and Device ciencies Definitions and Procedures for Recording, Evaluating, | 0.5 |
|---|---|---|
| | ow-Up, and Reporting in Medical Device Studies | |
| | 0.5.2. Definition of SAE, SADE, and USADE | |
| | 0.5.3. Definition of Device Deficiency | 86 |
| 1 | 0.5.4. Recording/Reporting and Follow-Up of Medical Device Deficiencies | 86 |
| 1 | 0.5.5. Reporting of SAEs | 88 |
| 1 | 0.5.6. Reporting of SADEs | 88 |
| 10.6. A | ppendix 6: Alternative Measures During Public Emergencies | 89 |
| 1 | 0.6.1. Telehealth Visits | 89 |
| | ppendix 7: Criteria for Allowing Inclusion of Participants With Chronic le HIV, HCV, or HBV Infection | 90 |
| 10.8. A | ppendix 8: Abbreviations | 91 |
| 11. REFERE | NCES | 94 |
| | LIST OF TABLES | |
| Table 1. | Vaccine Administration Group | 31 |
| Table 2. | Grading Scale for Local Reactions | 43 |
| Table 3. | Grading Scale for Systemic Events | 44 |
| Table 4. | Ranges for Fever | 45 |
| Table 5. | Analysis Sets | 61 |
| Table 6. | Primary Endpoint Analyses | 63 |
| Table 7. | Secondary Endpoint Analyses | 64 |
| Table 8. | Exploratory Endpoint Analyses | 64 |
| Table 9. | Sample Size Determination | 65 |

#### 1. PROTOCOL SUMMARY

## 1.1. Synopsis

**Brief Title:** Safety and Immunogenicity of RSVpreF Coadministered With SIIV in Adults ≥65 Years of Age

#### Rationale

Annual seasonal influenza vaccination is recommended in a number of countries around the world to prevent influenza in children and adults. Older adults, particularly those with medical comorbidities, are at increased risk of influenza morbidity and mortality and are recommended to receive high-dose or adjuvanted influenza vaccine formulations. RSV and influenza are both typically seasonal diseases, with peaks during winter in temperate climates. Therefore, it is a possibility that RSVpreF may be given at the same time as seasonal influenza vaccine.

The purpose of this study is to assess the safety and immunogenicity of RSVpreF when coadministered with SIIV compared to sequential administration of the vaccines when given 1 month apart (SIIV followed by RSVpreF). Additionally, the study will contribute data supporting the development of RSVpreF as a prophylactic vaccine against RSV disease in infants through maternal immunization and in older adults through active vaccination.

## Objectives, Endpoints, and Estimands

| Objectives | Endpoints | Estimands |
|---|---|---|
| Primary Safety | | |
| To evaluate the safety profiles of RSVpreF when coadministered with SIIV (RSVpreF + SIIV) or when administered 1 month after SIIV. | <ul> <li>Local reactions (redness, swelling, and pain at the injection site) self-reported on e-diaries for 7 days after vaccination.</li> <li>Systemic events (fever, fatigue, headache, nausea, vomiting, diarrhea, muscle pain, and joint pain) self-reported on e-diaries for 7 days after vaccination.</li> <li>AEs.</li> <li>SAEs.</li> </ul> | In participants receiving 1 dose of study intervention and having safety follow-up after vaccination from each vaccine group: • The percentage of participants reporting prompted local reactions and systemic events within 7 days after vaccination with RSVpreF or placebo. • The percentage of participants reporting AEs and SAEs within 1 month after each vaccination. |

| Objectives | Endpoints | Estimands |
|---|---|---|
| Primary RSV Immunogenicity | | |
| To demonstrate that the immune responses elicited by RSVpreF when coadministered with SIIV (RSVpreF + SIIV) are noninferior to those elicited by RSVpreF alone when administered 1 month after SIIV. | RSV A and RSV B NTs. | In participants in compliance with the key protocol criteria (evaluable participants): • GMR of NTs at 1 month after vaccination with RSVpreF for each RSV subfamily (A or B) in RSVpreF + SIIV to RSVpreF alone (sequential-administration group). |
| Primary SIIV Immunogenicity | y | |
| To demonstrate that the immune responses elicited by SIIV when coadministered with RSVpreF (RSVpreF + SIIV) are noninferior to those elicited by SIIV alone. | <ul> <li>Strain-specific HAI titers.</li> <li>H3N2-neutralizing antibody titers (if interpretable H3N2-HAI titers cannot be obtained).</li> </ul> | In participants in compliance with the key protocol criteria (evaluable participants): • GMR of the strain-specific HAI (or H3N2-neutralizing antibody) titers 1 month after vaccination with SIIV in the coadministration group to the corresponding HAI (or H3N2-neutralizing antibody) titers in the sequential-administration group. |
| Secondary RSV Immunogenic | Secondary RSV Immunogenicity | |
| To describe immune responses elicited by RSVpreF when coadministered with SIIV or when administered alone. | RSV A and RSV B NTs. | In participants in compliance with the key protocol criteria (evaluable participants) from each vaccine group: Geometric mean of the NTs for RSV A and RSV B before vaccination and at each applicable visit after vaccination with RSVpreF. GMFR of the NTs for RSV A and RSV B before vaccination and at each applicable visit after vaccination with RSVpreF. |
| Secondary SIIV Immunogenicity | | |
| To describe immune responses elicited by SIIV when coadministered with RSVpreF or when administered alone. | <ul> <li>Strain-specific HAI titers.</li> <li>H3N2-neutralizing antibody titers (if interpretable H3N2-HAI titers cannot be obtained).</li> </ul> | In participants in compliance with the key protocol criteria (evaluable participants) from each vaccine group: • GMTs before vaccination and 1 month after vaccination with SIIV. |

| Objectives | Endpoints | Estimands |
|---|---|---|
| | | GMFR of strain-specific HAI titers (or H3N2-neutralizing antibody titers if interpretable H3N2-HAI titers cannot be obtained) before vaccination and 1 month after vaccination with SIIV. |
| CCI | | |
| Exploratory SIIV Immunogen | icity | |
| To further describe immune responses elicited by SIIV when coadministered with RSVpreF or when administered alone. | <ul> <li>Strain-specific HAI titers.</li> <li>H3N2-neutralizing antibody titers (if interpretable H3N2-HAI titers cannot be obtained).</li> </ul> | |

## **Overall Design**

## **Brief Summary**

This Phase 3, multicenter, parallel-group, placebo-controlled, randomized, double-blind study will be conducted in Australia and/or another southern hemisphere country.

Healthy adults ≥65 years of age will be randomized 1:1 to either the coadministration group (RSVpreF + SIIV)/placebo or the sequential-administration group (placebo + SIIV)/RSVpreF.

There are 3 scheduled study visits each 1 month apart. To assess immunogenicity, blood will be collected prior to vaccination at Visit 1 and Visit 2, and at Visit 3.

Local reactions at the RSVpreF or placebo injection site (left deltoid) and systemic events occurring within 7 days after each vaccination will be recorded in an e-diary device or smartphone app.

AEs and SAEs will be collected from the signing of informed consent through study completion (Visit 3).

#### **Number of Participants**

Approximately 1400 healthy, older adults will be enrolled in the study.

## **Intervention Groups and Duration**

There will be 2 study groups:

Group 1 (coadministration):

• Visit 1: (RSVpreF + SIIV)

• Visit 2: placebo

Group 2 (sequential administration):

• Visit 1: (placebo + SIIV)

• Visit 2: RSVpreF

Each participant will participate in the study for approximately 2 months. Based on an estimated 2-month enrollment period, the study duration will be approximately 4 months.

#### **Statistical Methods**

GMRs of RSV NTs in the coadministration group to the sequential-administration group for RSV A and RSV B at 1 month after vaccination with RSVpreF will be provided along with associated 2-sided 95% CIs. GMRs of strain-specific HAI titers in the coadministration group to the sequential-administration group at 1 month after vaccination with SIIV will be provided along with associated 2-sided 95% CIs. Using a 1.5-fold margin, noninferiority will be declared if the lower bound of the 2-sided 95% CI for each GMR is greater than 0.667 for all SIIV strains and for both RSV A and RSV B.

The primary safety objective will be evaluated by descriptive summary statistics for local reactions, systemic events, AEs, and SAEs after each vaccination for each vaccine group. A 3-tier approach will be used to summarize AEs.

# 1.2. Study Design Schema

| Healthy Adults<br>≥65 Years of Age | | Visit | 1 | Visit 2<br>28-35 Days after Visit 1 | Visit 3 28-35 Days after Visit 2 |
|---|---|---|---|---|---|
| | | Day 1<br>Vaccination 1 | | Month 1<br>Vaccination 2 | Month 2<br>Follow-Up |
| Study Group (n) | | Injectio<br>delto<br><b>Left</b> | | Injection site:<br>deltoid<br><b>Left</b> | |
| <b>Group 1</b> 700 | Coadministration RSVpreF + SIIV/placebo | RSVpreF | SIIV | Placebo | • |
| <b>Group 2</b> 700 | Sequential<br>administration<br>Placebo +<br>SIIV/RSVpreF | Placebo | SIIV | RSVpreF | • |
| | Safety assessments: reactogenicity, AEs/SAEs | | | | |
| 30-mL blood draw 120 µg RSVpreF (blinded administration) SIIV (unblinded administration) Placebo (blinded administration) | | | | | |

### 1.3. Schedule of Activities

The SoA table provides an overview of the protocol visits and procedures. Refer to Study Assessments and Procedures in Section 8 for detailed information on each procedure and assessment required for compliance with the protocol. The investigator may schedule visits (unplanned visits) in addition to those listed in the SoA table, to conduct evaluations or assessments required in order to protect the well-being of the participant.

## **Schedule of Activities**

| Visit Identifier | Visit 1 | Visit 2 | Visit 3 |
|---|---|---|---|
| Visit Description | Day 1 | Month 1 | Month 2 |
| Visit Window | Vaccination 1 | Vaccination 2<br>28-35 Days<br>after Visit 1 | 28-35 Days<br>after Visit 2 |
| Obtain informed consent | X | | |
| Obtain participant number via IRT | X | | |
| Obtain demography and significant medical history data | X | | |
| Record current/former tobacco usage | X | | |
| Perform clinical assessment (and physical examination if deemed necessary) | X | | |
| Record nonstudy vaccinations, review concomitant medication use | X | X | X |
| Review inclusion and exclusion criteria and confirm eligibility | X | | |
| Obtain participant's temperature | X | X | |
| Review temporary delay criteria | X | X | |
| Obtain blood sample for antibody assessment (~30 mL) | Xa | Xa | X |
| Obtain randomization number and kit assignment from IRT | X | | |
| Explain/review participant communication methods, assist with downloading the e-diary application, or issue provisioned e-diary device, if required. | X | | |
| Provide e-diary training, issue thermometer and measuring device | X | X <sup>b</sup> | |
| Administer SIIV in right deltoid muscle | X | | |
| Administer study intervention in left deltoid muscle | X | X | |
| Discuss contraceptive use (as appropriate) | X | X | |
| Issue ECC and explain its purpose and use | X | $X^{b}$ | |
| Postvaccination observation (30 minutes) and immediate reaction assessment | X | X | |
| Review e-diary data,(daily during the 7 days after vaccination) | X | X | |
| Review e-diary for ongoing events and stop dates, collect e-diary <sup>c</sup> | | X | X |
| Record AEs/SAEs and stop dates for previously reported events. | X | X | X |

- a. Blood sample must be collected before vaccination.
- b. Issue replacement thermometer, measuring device, and ECC, only if required
- c. Collect provisioned e-diaries at Visit 3 only.

#### 2. INTRODUCTION

RSV is a major cause of respiratory infection in all ages, which can result in severe illness in both infants and older adults. There are 2 antigenic variants of RSV: subgroups A (RSV A) and B (RSV B) that cocirculate. Like influenza, RSV infection follows a seasonal pattern, causing yearly wintertime epidemics in temperate climates, usually between late autumn and early spring. In tropical climates, the outbreaks are generally associated with rainy seasons but are more unpredictable and frequently continuous. Due to the COVID-19 pandemic, which spread worldwide in 2020 and 2021, the seasonality of several pathogens, including RSV, has been disrupted and the shift of peak incidence has been observed in a majority of geographies. Therefore the RSV season is less predictable with respect to onset and duration.

Adults >60 years of age have an increased risk of RSV infection, which can trigger exacerbations of underlying comorbid conditions, such as COPD and CHF. RSV infection has been associated with up to 22% of acute COPD exacerbations in prospective cohort studies and 11% of wintertime hospitalizations for COPD exacerbations. 4 Current epidemiology shows that RSV is responsible for approximately 177,000 hospitalizations and 14,000 deaths annually in US adults 65 years of age and older. Morbidity is significant among adults hospitalized with RSV disease, with 18% requiring intensive care, 31% needing home health services at discharge, and 26% dying within 1 year of hospitalization.<sup>6</sup> In the US, RSV disease incidence rates in older adults are approximately half those of influenza, with variation year to year. Incidence rates and risk for severe complications from RSV infection are higher among immunocompromised adults and those with chronic conditions (eg, cardiopulmonary or renal disease, hematological malignancies, receipt of chemotherapy, or HIV infection).<sup>8,9</sup> However, the burden of adult RSV disease could be underestimated since testing for RSV is less common in older adults than in children. RSV disease in adults is also difficult to diagnose based on clinical signs and symptoms alone, and, prior to the broader use of more sensitive detection methods, laboratory confirmation of RSV in adults was challenging because of low levels of virus shedding.<sup>4</sup>

RSV disease management in adults is limited to supportive measures, such as hydration and oxygenation. Aerosolized ribavirin has limited evidence of effectiveness and is predominantly restricted to severely immunocompromised hospitalized patients because of inconvenient administration, teratogenicity, anemia concerns, and high cost. Prevention of RSV disease via active immunization has the potential to make a significant impact in this population, therefore making vaccine development a high priority. <sup>9,10</sup>

## 2.1. Study Rationale

Annual seasonal influenza vaccination is recommended in a number of countries around the world to prevent influenza in children and adults. Older adults, particularly those with medical comorbidities, are at increased risk of influenza morbidity and mortality and are recommended to receive high-dose or adjuvanted influenza vaccine formulations. RSV and influenza are both typically seasonal diseases, with peaks during winter in temperate climates. Therefore, it is a possibility that RSV preF may be given at the same time as seasonal influenza vaccine.

• The purpose of this study is to assess the safety and immunogenicity of RSVpreF when coadministered with SIIV, compared to sequential administration of the vaccines when given 1 month apart (SIIV followed by RSVpreF). Additionally, the study will contribute data supporting the development of RSVpreF as a prophylactic vaccine against RSV disease in infants through maternal immunization and in older adults through preventive vaccination.

## 2.2. Background

The vaccine under evaluation in this study is a bivalent RSV prefusion F subunit vaccine developed by Pfizer. The RSV F glycoprotein facilitates fusion of the virion and host cell membrane through a dramatic transition from an unstable but highly immunogenic prefusion conformation to the more stable postfusion state. Preclinical studies show that prefusion F elicits much higher neutralizing antibody titers than postfusion F and that the most potent neutralizing antibodies from postinfection human sera target the prefusion form. RSVpreF is composed of engineered, stabilized, trimeric, prefusion F glycoproteins matching the A and B subgroups to help ensure the broadest coverage against RSV illness.

Pfizer's RSV stabilized prefusion F subunit vaccine (RSVpreF) is a prophylactic vaccine that is being developed for 2 indications:

- Older Adult: Prevention of RSV-associated LRTI in adults 60 years of age and older via active immunization.
- Maternal: Prevention of LRTI-RSV in infants by active immunization of pregnant women.

## 2.2.1. Clinical Overview

#### **Adult Program Studies**

The older adult program includes 2 Phase 1/2 studies, the human challenge study, and 2 Phase 3 studies.

- In the Phase 1/2 C3671001 study, 1233 healthy adults 18 through 49 and 50 through 85 years of age received the 3 dose levels of RSVpreF (60 μg, 120 μg, and 240 μg), with or without Al(OH)3, or placebo, administered with or without concomitant flu vaccine. The results have shown the vaccine was well tolerated and immunogenic in both age groups. RSVpreF elicited robust neutralizing responses against RSV A and RSV B 1 month after vaccination for both age groups across all vaccine dose levels and formulations and remained high through the 12 months after vaccination. In 616 vaccinated participants in the 50 to 85 years age group, RSV 50% NT GMFRs were high across all arms ranging from 9 to 13 from before vaccination to 1 month after vaccination and from 3 to 4 from before vaccination to 12 months after vaccination for RSV A and RSV B. When RSVpreF was coadministered with SIIV, trends in immune responses to RSVpreF were inconsistent depending on dose level and formulation. Immune responses to SIIV trended lower when coadministered with RSVpreF for both age groups, but the impact was less in the 65 to 85 years age group, compared to the 18 through 49 year age group. RSVpreF was safe and well tolerated when administered alone or with SIIV, with no major differences observed across all dose levels and formulations. Most reported local reactions or systemic events were mild or moderate in severity. Proportions of participants reporting AEs were generally similar across RSVpreF groups, and no SAEs were considered related to the study intervention.
- The Phase 1/2 C3671002 study in 313 older adults 65 to 85 years of age examined 3 dose levels of RSVpreF with Al(OH)<sub>3</sub> (60 μg, 120 μg, and 240 μg), formulated with or without CpG adjuvant, given as a single dose with concomitant SIIV or in a 2-dose regimen administered 2 months apart. All RSVpreF doses and formulations elicited high RSV A and RSV B neutralizing antibody GMTs 1 month after vaccination (GMFRs ranging from 4.8 to 11.6 and 4.5 to 14.1, respectively). CpG-containing formulations did not further increase neutralizing GMTs compared to RSVpreF with or without Al(OH)<sub>3</sub>. GMTs in all groups declined but remained higher than baseline (before vaccination) and placebo (SIIV only) at 12 months after vaccination (GMFRs ranging from 2.1 to 3.5 and 2.2 to 4.3, respectively). No increase in GMTs was observed 1 month after Vaccination 2 (GMFR of 0.9). All doses and formulations were safe and well tolerated. Immune responses to SIIV demonstrated by HAI titers and H3N2-neutralizing titers were similar or trended slightly lower in RSVpreF groups (coadministered with SIIV) compared to the placebo group (received SIIV only), and rates of seroprotection and seroconversion 1 month after SIIV administration were generally similar.
- A Phase 2a, randomized, double-blind, placebo-controlled study to evaluate the safety, immunogenicity, and efficacy of RSVpreF in a virus challenge model in healthy adults (NCT04785612) has been conducted in 70 healthy participants 18 to 50 years of age. Participants received a single dose of either 120 μg RSVpreF or placebo, and 4 weeks later underwent intranasal challenge with RSV A Memphis 37b virus. The immunogenicity and efficacy of RSVpreF vaccination on virus replication, clinical symptoms, and incidence of symptomatic RSV infection were evaluated. The primary analysis of the human challenge study showed that the 120-μg dose of RSVpreF is well tolerated and has an acceptable safety profile. The study has demonstrated 100% efficacy

of RSVpreF against RT-PCR-confirmed symptomatic respiratory infection in a mild-to-moderate disease model.

- Study C3671014 is a completed Phase 3, multicenter, parallel-group, placebo-controlled, randomized, double-blind lot consistency study in a population of up to 1000 healthy adults 18 to ≤49 years of age. The study examined the immune response and the safety and tolerability profiles across 3 manufactured lots of RSVpreF when administered as a single 120-μg dose to healthy adults. The primary analyses showed that the ratio of neutralizing GMTs for each of the 3 manufactured RSVpreF lots, 1 month after vaccination are equivalent, and that the 120-μg dose of RSVpreF is well tolerated and has an acceptable safety profile.
- Study C3671013 is an ongoing Phase 3, multicenter, randomized, double-blind, placebo-controlled study to assess the safety, immunogenicity, and efficacy of RSVpreF in the prevention of RSV-associated LRTI in adults 60 years of age and older. Both healthy adults and adults with stable chronic cardiopulmonary conditions will be included. Approximately 10% of participants with stable chronic cardiopulmonary conditions, such as COPD, asthma, or CHF, will be enrolled. Up to 45,000 participants will be randomized to receive RSVpreF or placebo in a 1:1 ratio. This is an event-driven study with a target of 59 first episodes of evaluable RSV-associated LRTI cases.

## **Maternal Program Studies**

The maternal program includes ongoing Phase 2b and 3 studies in pregnant women and a completed Phase 2b study in nonpregnant women. The Phase 3 lot consistency study C3671014 described under the adult program studies will contribute data to support the maternal immunization program. Analyses and ongoing safety reviews in each of these studies have demonstrated that RSVpreF has a good safety and tolerability profile and no safety signals were identified. Further details are described in the IB.

## 2.3. Benefit/Risk Assessment

More detailed information about the known and expected benefits and risks and reasonably expected AEs of RSVpreF may be found in the IB, which is the SRSD for this study.

The SRSD for the SIIV will be the product information for the country where the vaccine was procured.

# 2.3.1. Risk Assessment

| Potential Risk of Clinical<br>Significance | Summary of Data/Rationale for Risk | Mitigation Strategy |
|---|---|---|
| Study Intervention(s): RSVpreF | | |
| Local reactions and systemic events to the vaccine may occur (injection site redness, injection site swelling, and injection site pain; fever, fatigue, headache, nausea, vomiting, diarrhea, muscle pain, and joint pain) following vaccination. | These are common adverse reactions seen with other vaccines <sup>13</sup> as well as RSVpreF. The most common events reported in Study C3671001 were mild-to-moderate pain at the injection site, fatigue, headache, and muscle pain. | The study employs the use of a reactogenicity e-diary, which allows the investigator to monitor local reactions and systemic events in real time through an electronic portal. Severe reactions will require an unscheduled telephone call, and if required a clinic visit, to be conducted per the protocol. All study participants will be observed for at least 30 minutes after vaccination. |
| Safety profile of a novel vaccine close to being, but not yet fully, characterized. | Data available from completed and ongoing studies showed a low incidence of severe or serious events and no clinically concerning safety observations. The vaccine appears to be safe and well tolerated across the safety population and within demographic subgroups based on age, sex, and race/ethnicity. | <ul> <li>Assessments of AEs and SAEs will be collected and reviewed throughout the study.</li> <li>All participants will be observed for at least 30 minutes after vaccination.</li> </ul> |
| Theoretical risk for RSV enhancement. | RSVpreF is being evaluated in ongoing clinical studies. Pfizer's immunization approach circumvents the risk of vaccine-mediated disease enhancement that was observed in the 1960s following direct immunization of RSV-naive infants with an FI-RSV. FI-RSV elicited a predominantly nonneutralizing antibody response and a Th2-biased cell-mediated response, both of which are considered potential contributing factors to disease enhancement. During preclinical studies, in a standard cotton rat infectious RSV challenge model, FI-RSV showed pathological signs of causing disease enhancement, and the current Pfizer vaccine candidate, RSVpreF, did not. Most important, RSV vaccine—mediated disease enhancement has not been reported in RSV-experienced individuals after vaccination with any RSV vaccine candidate. Because older adults are universally RSV-experienced, they are not considered at risk for a disease-enhancing immune response to the vaccine or a potential exacerbation of an infection. | Assessments of AEs and SAEs will be collected and reviewed throughout the study. |

| Potential Risk of Clinical<br>Significance | Summary of Data/Rationale for Risk | Mitigation Strategy |
|---|---|---|
| Concomitant Vaccine: SIIV | | |
| The relevant key risks associated with SIIV include injection site pain, fatigue, headache, redness at the injection site, joint pain, muscle pain, and diarrhea. <sup>14</sup> | The risks are based on the SIIV product information for the country where the vaccine was procured. | Eligibility criteria have been selected to ensure that only appropriate participants are included in the study, including those who may have contraindications to SIIV components/administration (see Section 5). |
| Coadministration of<br>RSVpreF with SIIV may<br>enhance local and<br>systemic reactions. | RSVpreF has already been coadministered with SIIV in Studies C3671001 and C3671002 including older adult populations. There was no evidence of enhancement of local reactions and systemic events associated with concomitant administration in these studies and no safety concerns. | E-diary and AE data will be monitored by the investigator (or designee) and sponsor. Participants who develop exclusionary conditions during study conduct or participants with significant reactions after Visit 1 vaccinations or AEs considered by the investigator to present increased risk to the participant if he/she received additional study vaccinations may be excluded from further vaccinations. |
| Coadministration of RSVpreF with SIIV may impact the immune response to SIIV. In Study C3671001, immune responses to SIIV trended lower when coadministered with RSVpreF, while in Study C3671002, immune responses to SIIV were similar or slightly lower, and HAI seroprotection and seroconversion rates remained similar. | | Based on Phase 1/2 data, this risk is considered low, given comparable seroprotection rates observed in the older adult population; however, influenza cases will be collected as AEs or SAEs. |
| Study Procedures | | |
| Venipuncture will be performed during the study. | There is the risk of bleeding, bruising, hematoma formation, and infection at the venipuncture site. | Only appropriately qualified personnel will obtain the blood draw. |
| Participants will be required to attend healthcare facilities during the global SARS-CoV-2 pandemic. | Without appropriate social distancing and PPE, there is a potential for increased exposure to SARS-CoV-2. | <ul> <li>Pfizer will work with sites to<br/>ensure appropriate COVID-19<br/>prevention strategies.</li> <li>Cases of COVID-19 will be<br/>reported as AEs or SAEs.</li> </ul> |

#### 2.3.2. Benefit Assessment

Benefit considerations may include:

- Potential benefit of receiving study intervention that may have clinical utility in the future.
- Contributing to the process of developing new therapies in an area of unmet need.
- Medical evaluations/assessments associated with study procedures.
- Receipt of a licensed influenza vaccine.

#### 2.3.3. Overall Benefit/Risk Conclusion

Taking into account the measures to minimize risk to study participants, the potential risks identified in association with RSVpreF are justified by the anticipated benefits that may be afforded to study participants who may be at risk of RSV.

## 3. OBJECTIVES, ENDPOINTS, AND ESTIMANDS

| Objectives | Endpoints | Estimands |
|---|---|---|
| Primary Safety | - | |
| To evaluate the safety profiles of RSVpreF when coadministered with SIIV (RSVpreF + SIIV) or administered 1 month after SIIV. | <ul> <li>Local reactions (redness, swelling, and pain at the injection site) self-reported on e-diaries for 7 days after vaccination.</li> <li>Systemic events (fever, fatigue, headache, nausea, vomiting, diarrhea, muscle pain, and joint pain) self-reported on e-diaries for 7 days after vaccination.</li> <li>AEs.</li> <li>SAEs.</li> </ul> | In participants receiving 1 dose of study intervention and having safety follow-up after vaccination from each vaccine group: The percentage of participants reporting prompted local reactions and systemic events within 7 days after vaccination with RSVpreF or placebo. The percentage of participants reporting AEs and SAEs within 1 month after each vaccination. |
| Primary RSV Immunogenicity | y | |
| To demonstrate that the immune responses elicited by RSVpreF when coadministered with SIIV (RSVpreF + SIIV) are noninferior to those elicited by RSVpreF alone when administered 1 month after SIIV. | RSV A and RSV B NTs. | In participants in compliance with the key protocol criteria (evaluable participants): • GMR of NTs at 1 month after vaccination with RSVpreF for each RSV subfamily (A or B) in RSVpreF + SIIV to RSVpreF alone (sequential-administration group). |

| Objectives | Endpoints | Estimands |
|---|---|---|
| Primary SIIV Immunogenicity | | |
| To demonstrate that the immune responses elicited by SIIV when coadministered with RSVpreF (RSVpreF + SIIV) are noninferior to those elicited by SIIV alone. | <ul> <li>Strain-specific HAI titers.</li> <li>H3N2-neutralizing antibody titers (if interpretable H3N2-HAI titers cannot be obtained).</li> </ul> | In participants in compliance with the key protocol criteria (evaluable participants): • GMR of the strain-specific HAI (or H3N2-neutralizing antibody) titers 1 month after vaccination with SIIV in the coadministration group to the corresponding HAI (or H3N2-neutralizing antibody) titers in the sequential-administration group |
| Secondary RSV Immunogenic | ity | |
| To describe immune responses elicited by RSVpreF when coadministered with SIIV or when administered alone. | RSV A and RSV B NTs. | In participants in compliance with the key protocol criteria (evaluable participants) from each vaccine group: Geometric mean of the NTs for RSV A and RSV B before vaccination and at each applicable visit after vaccination with RSVpreF. GMFR of the NTs for RSV A and RSV B before vaccination and at each applicable visit after vaccination with RSVpreF. |
| Secondary SIIV Immunogenic | ity | |
| To describe immune responses elicited by SIIV when coadministered with RSVpreF or when administered alone. | Strain-specific HAI titers. H3N2-neutralizing antibody titers (if interpretable H3N2-HAI titers cannot be obtained). | <ul> <li>In participants in compliance with the key protocol criteria (evaluable participants) from each vaccine group:</li> <li>GMTs before vaccination and 1 month after vaccination with SIIV.</li> <li>GMFR of strain-specific HAI titers (or H3N2-neutralizing antibody titers if interpretable H3N2-HAI titers cannot be obtained) before vaccination and 1 month after vaccination with SIIV.</li> </ul> |

| Objectives | Endpoints | Estimands |
|---|---|---|
| CCI | | |
| <b>Exploratory SIIV Immunogen</b> | icity | |
| To further describe immune responses elicited by SIIV when coadministered with RSVpreF or when administered alone. | <ul> <li>Strain-specific HAI titers.</li> <li>H3N2-neutralizing antibody titers (if interpretable H3N2-HAI titers cannot be obtained).</li> </ul> | |

#### 4. STUDY DESIGN

## 4.1. Overall Design

This Phase 3, multicenter, parallel-group, placebo-controlled, randomized, double-blind study will be conducted in Australia and/or another southern hemisphere country.

Healthy adults >65 years of age will be randomized 1:1 to either the coadministration group (RSVpreF + SIIV)/placebo or the sequential-administration group (placebo + SIIV)/RSVpreF. This study design intends to use a single lot of SIIV that is specifically indicated for use in adults ≥65 years of age; however, the SIIV ultimately used may be determined by supply availability.

There are 3 scheduled study visits each 1 month apart. To assess immunogenicity, 30 mL blood will be collected prior to vaccination at Visit 1 and Visit 2, and at Visit 3.

Local reactions (redness, swelling, and pain at the injection site) occurring at the RSVpreF or placebo injection site (left deltoid) and systemic events (fever, headache, fatigue, nausea, vomiting, diarrhea, muscle pain, and joint pain) occurring within 7 days after each vaccination visit (Visit 1 and Visit 2) will be prompted for and collected daily by the participant in an e-diary device or smartphone app. SIIV injection site reactions will not be routinely collected in the e-diary.

AEs and SAEs will be collected from the signing of informed consent through Visit 3.

#### **Number of Participants**

Approximately 1400 participants (700 per group) will be enrolled in the study. Participants who withdraw or are withdrawn from the study after randomization will not be replaced, regardless of the reason for withdrawal.

## **Intervention Groups and Duration**

There will be 2 study groups:

Group 1 (coadministration):

• Visit 1: (RSVpreF + SIIV)

• Visit 2: placebo

Group 2 (sequential administration):

• Visit 1: (placebo + SIIV)

• Visit 2: RSVpreF

Each participant will participate in the study for approximately 2 months. Based on an estimated 2-month enrollment period, the total study duration will be approximately 4 months.

## 4.2. Scientific Rationale for Study Design

See Section 2.1.

## 4.2.1. Choice of Contraception/Barrier Requirements

There is no suspicion of human teratogenicity based on the available reproductive toxicity data; however, human reproductive safety data are limited, and a Phase 3 study of RSVpreF in pregnant women is ongoing. Therefore, the use of a highly effective method of contraception is required (see Section 10.3, Appendix 3).

#### 4.3. Justification for Dose

The final dose and formulation of RSVpreF selected for use in this study is based on the safety and immunogenicity data from 3 Phase 1/2 studies and the efficacy evaluation in the human challenge study.

- The FIH study in adults 18 through 85 years of age evaluated the safety, tolerability, and immunogenicity of 3 escalating RSVpreF dose levels of 60 μg, 120 μg, and 240 μg, with or without Al(OH)3, when administered alone or concomitantly with SIIV (Study C3671001).
- A study in older adults 65 through 85 years of age evaluated the safety, tolerability, and immunogenicity of 60 μg, 120 μg, and 240 μg RSVpreF doses formulated with Al(OH)3 or a CpG/Al(OH)3 adjuvant, or 240 μg RSVpreF with RSV antigens alone, when administered concomitantly with SIIV (Study C3671002).

• A study in healthy adults 18 through 50 years of age evaluated the safety, immunogenicity, and efficacy of 120 μg RSVpreF in a virus challenge model (NCT04785612).

Based on the Phase 1/2 studies (C3671001 and C3671002), no substantial differences were observed between the immunogenicity or reactogenicity of the 120-µg and 240-µg dose levels or of formulations with and without Al(OH)3 or CpG/Al(OH)3. Therefore, the 120-µg without-Al(OH)3 formulation was chosen for the human challenge study. The acceptable reactogenicity and safety profile along with the high efficacy demonstrated in the primarily-upper-respiratory-tract and mild-to-moderate disease human challenge model led to the selection of a 120-µg dose for the RSV Phase 3 studies.

## 4.4. End of Study Definition

The end of the study is defined as the date of the last visit of the last participant in the study.

A participant is considered to have completed the study when she/he has completed all study visits.

#### 5. STUDY POPULATION

This study can fulfill its objectives only if appropriate participants are enrolled, including participants across diverse and representative racial and ethnic backgrounds. Use of a prescreener for study recruitment purposes will include collection of information that reflects the enrollment of a diverse participant population including, where permitted under local regulations, age, sex, race, and ethnicity. The following eligibility criteria are designed to select participants for whom participation in the study is considered appropriate. All relevant medical and nonmedical conditions should be taken into consideration when deciding whether a particular participant is suitable for this protocol.

Prospective approval of protocol deviations to recruitment and enrollment criteria, also known as protocol waivers or exemptions, is not permitted.

#### 5.1. Inclusion Criteria

Participants are eligible to be included in the study only if all the following criteria apply:

## Age and Sex:

1. Male and female participants  $\geq$ 65 years of age at the time of consent.

Refer to Appendix 3 for reproductive criteria for male (Section 10.3.1) and female (Section 10.3.2) participants.

## Type of Participant and Disease Characteristics:

- 2. Participants who are willing and able to comply with scheduled visits, laboratory tests, lifestyle considerations, and other study procedures, including daily completion of the e-diary for 7 days after each study vaccination.
- 3. Healthy participants who are determined by medical history, physical examination (if required), and clinical judgment of the investigator to be eligible for inclusion in the study.

Note: Healthy participants with preexisting stable disease, defined as disease not requiring significant change in therapy or hospitalization for worsening disease during the 6 weeks before enrollment, can be included. Specific criteria for participants with known stable infection with HIV, HCV, or HBV can be found in Section 10.7, Appendix 7.

#### **Informed Consent:**

4. Capable of giving signed informed consent as described in Appendix 1, which includes compliance with the requirements and restrictions listed in the ICD and in this protocol.

## 5.2. Exclusion Criteria

Participants are excluded from the study if any of the following criteria apply:

#### **Medical Conditions:**

- 1. Bleeding diathesis or condition associated with prolonged bleeding time that may contraindicate IM injection.
- 2. History of severe adverse reaction associated with a vaccine and/or severe allergic reaction (eg, anaphylaxis) to any component of the study intervention or any related vaccine.
- 3. Allergy to egg proteins (egg or egg products) or chicken proteins.
- 4. History of Guillain-Barré syndrome.
- 5. Serious chronic disorder, including metastatic malignancy, end-stage renal disease with or without dialysis, clinically unstable cardiac disease, or any other disorder that, in the investigator's opinion, excludes the participant from participating in the study.
- 6. Immunocompromised individuals with known or suspected immunodeficiency, as determined by history and/or laboratory/physical examination.
- 7. Other medical or psychiatric condition, including recent (within the past year) or active suicidal ideation/behavior, or laboratory abnormality that may increase the risk of study participation or, in the investigator's judgment, make the participant inappropriate for the study.

## **Prior/Concomitant Therapy:**

- 8. Previous vaccination with any licensed or investigational RSV vaccine at any time prior to enrollment, or planned receipt throughout the study of nonstudy RSV vaccine.
- 9. Previous vaccination with any influenza vaccine within 6 months before study intervention administration, or planned receipt of any nonstudy licensed or investigational influenza vaccine during study participation.
- 10. Receipt of any blood/plasma products or immunoglobulin, from 60 days before study intervention administration, or planned receipt throughout the study.
- 11. Individuals who receive chronic treatment with immunosuppressive therapy, including cytotoxic agents, monoclonal antibodies, systemic corticosteroids, or radiotherapy, eg, for cancer or an autoimmune disease, from 60 days before study intervention administration or planned receipt throughout the study. If systemic corticosteroids (<20 mg/day of prednisone or equivalent) have been administered short term (<14 days) for treatment of an acute illness, participants should not be enrolled in the study until corticosteroid therapy has been discontinued for at least 28 days before study intervention administration. Inhaled/nebulized, intraarticular, intrabursal, or topical (skin or eyes) corticosteroid use is permitted.

Note: Participants with COPD or asthma can be enrolled if chronic corticosteroids do not exceed a dose equivalent to 10 mg/day of prednisone.

- 12. Current alcohol abuse or illicit drug use.
- 13. Current use of any prohibited concomitant medication(s) or those unwilling/unable to use a permitted concomitant medication(s). Refer to Section 6.10.

## **Prior/Concurrent Clinical Study Experience:**

14. Participation in other studies involving investigational product(s) within 28 days prior to consent and/or during study participation.

#### **Other Exclusions:**

15. Investigator site staff or Pfizer employees directly involved in the conduct of the study, site staff otherwise supervised by the investigator, and their respective family members.

## 5.3. Lifestyle Considerations

## **5.3.1.** Contraception

The investigator or his or her designee, in consultation with the participant, will confirm that the participant has selected an appropriate method of contraception for the individual participant from the permitted list of contraception methods (see Appendix 3, Section 10.3) and will confirm that the participant has been instructed in its consistent and correct use. At time points indicated in the SoA, the investigator or designee will inform the participant of the need to use highly effective contraception consistently and correctly and document the conversation and the participant's affirmation in the participant's chart (participants need to affirm their consistent and correct use of at least 1 of the selected methods of contraception) considering that their risk for pregnancy may have changed since the last visit. In addition, the investigator or designee will instruct the participant to call immediately if the selected contraception method is discontinued or if pregnancy is known or suspected in the participant or partner.

#### 5.4. Screen Failures

Screen failures are defined as participants who consent to participate in the clinical study but are not subsequently randomly assigned to study intervention. A minimal set of screen failure information is required to ensure transparent reporting of screen failure participants to meet the CONSORT publishing requirements and to respond to queries from regulatory authorities. Minimal information includes demography, screen failure details, eligibility criteria, and any SAE.

Individuals who do not meet the criteria for participation in this study (screen failure) may be rescreened under a new participant number.

# 5.5. Criteria for Temporarily Delaying Enrollment/Randomization/Administration of Study Intervention

The following conditions may allow a participant to be vaccinated once the conditions have resolved and the participant is otherwise eligible:

- Current febrile illness (body temperature ≥38°C [≥100.4°F]) or other acute illness within 48 hours before study intervention administration.
- Receipt of any inactivated vaccine, licensed COVID-19 vaccines, or COVID-19 vaccines authorized for temporary or emergency use within 14 days or any live vaccine within 28 days before study intervention administration.
- Receipt of short-term (<14 days) systemic corticosteroids. Study intervention administration should be delayed until systemic corticosteroid use has been discontinued for at least 28 days. Inhaled/nebulized, intra-articular, intrabursal, or topical (skin or eyes) corticosteroids are permitted.

## 6. STUDY INTERVENTION(S) AND CONCOMITANT THERAPY

Study intervention is defined as any investigational intervention(s), marketed product(s), placebo, medical device(s), or study procedure(s) intended to be administered to a study participant according to the study protocol.

For the purposes of this protocol, study intervention refers to RSVpreF and placebo (lyophilized cake containing excipients reconstituted in sterile water for injection).

Commercially available SIIV will be provided by the sponsor as a concomitant vaccine.

## 6.1. Study Intervention(s) Administered

## 6.1.1. Respiratory Syncytial Virus Stabilized Prefusion F Subunit Vaccine

| <b>Intervention Name</b> | RSVpreF |
|---|---|
| Туре | Vaccine |
| Dose Formulation | The active ingredients in RSVpreF are 2 stabilized RSV prefusion F antigens, in equal amounts from virus subgroups A and B, in a lyophilized dosage form for reconstitution. The RSV study intervention will be 120 µg of the RSV prefusion F antigen. The study intervention is supplied as a lyophilized white cake in a 2-mL glass vial, with a 13-mm lyophilization stopper, aluminum overseal, and flip-off cap. The study intervention will be reconstituted by a diluent consisting of sterile water in a PFS. The lyophilized cake contains excipients that, after reconstitution, will yield a solution as detailed in the IB. The fill volume of the study intervention vial and diluent PFS are designed such that the intended vaccine dose is delivered by injecting the entire contents of the syringe. |
| Dosage Level(s) | 120 μg RSVpreF by a single injection. |
| Route of<br>Administration | IM injection into the deltoid muscle of the LEFT arm. |
| Use | Experimental |
| Sourcing | RSVpreF will be provided by the sponsor to each study site. |
| Packaging and<br>Labeling | RSVpreF will be packaged within cartons labeled by Pfizer or its designee in accordance with current guidelines and applicable local and legal regulatory requirements. |

| <b>Intervention Name</b> | Placebo |
|---|---|
| Type | Placebo |
| Dose Formulation | The placebo is supplied as a lyophilized white cake in a 2-mL glass vial, with a 13-mm lyophilization stopper, aluminum overseal, and flip-off cap. It contains no active ingredients. The placebo will be reconstituted by a diluent consisting of sterile water in a PFS. The lyophilized cake contains excipients that, after reconstitution, will yield a volume matching RSVpreF. The fill volume of the placebo vial and diluent PFS are designed such that the intended vaccine dose is delivered by injecting the entire contents of the syringe. |

| <b>Intervention Name</b> | Placebo |
|---|---|
| Route of Administration | IM injection into the deltoid muscle of the LEFT arm. |
| Use | Placebo control |
| Sourcing | Placebo will be provided by the sponsor to each study site. |
| Packaging and<br>Labeling | The placebo will be packaged within cartons labeled by Pfizer or its designee in accordance with current guidelines and applicable local and legal regulatory requirements. |

#### 6.1.2. Concomitant Seasonal Inactivated Influenza Vaccine

Commercially available quadrivalent adjuvanted SIIV (if available), or an appropriate alternative SIIV for this older adult population, will be provided. Investigational sites will be notified which commercially available SIIV will be provided prior to the start of enrollment.

Pfizer will provide this vaccine; however, with approval by the sponsor, a site may independently procure the study-specific SIIV rather than receive shipment of SIIV from the sponsor. SIIV will be shipped and stored as per the commercial package insert and commercial label. Administration of SIIV will be recorded in the CRF and study records.

#### 6.2. Administration

RSVpreF and placebo will be prepared and administered by a blinded site staff member by injecting the entire contents of the syringe into the LEFT deltoid muscle.

SIIV will be prepared and administered by injecting the entire contents of the syringe into the deltoid muscle of the RIGHT arm. **No** blinding is required for the preparation or administration of SIIV.

Administration is summarized below.

**Table 1. Vaccine Administration Group** 

| Product Administered | | Visit 1 Vaccination 1 | Visit 2 Vaccination 2 |
|---|---|---|---|
| Group 1 Coadministration | Right deltoid muscle | SIIV | |
| | Left deltoid muscle | RSVpreF | Placebo |
| Group 2 Sequential Administration | Right deltoid muscle | SIIV | |
| | Left deltoid muscle | Placebo | RSVpreF |

Abbreviation: SIIV = seasonal inactivated influenza vaccine.

Administration of study interventions should be performed by an appropriately qualified, GCP-trained, and vaccine-experienced member of the study staff (eg, physician, nurse, physician's assistant, nurse practitioner, pharmacist, or medical assistant) as allowed by local, state, and institutional guidance.

Standard vaccination practices must be observed, and vaccine must not be injected into blood vessels. Appropriate medication and other supportive measures for management of an acute hypersensitivity reaction should be available in accordance with local guidelines for standard immunization practices.

Study intervention administration details will be recorded on the CRF and pharmacy/study records.

#### 6.3. Medical Devices

In this study, medical devices being deployed are for the reconstitution diluent for the study intervention. The study intervention supplies are provided in a kit that contains a vial of either RSVpreF or placebo lyophilized powder, a PFS containing sterile water, and a vial adapter. Instructions for their use are provided in the IPM.

Medical device deficiencies, including those resulting from malfunctions of the device, must be detected, documented, and reported by the study personnel throughout the study. Please refer to Section 8.3.9 for details.

#### 6.4. Preparation, Handling, Storage, and Accountability

- The investigator or designee must confirm appropriate temperature conditions have been maintained during transit for all study interventions received and any discrepancies are reported and resolved before use of the study intervention.
- Only participants enrolled in the study may receive study intervention and only authorized site staff may supply or administer study intervention. All study interventions must be stored in a secure, environmentally controlled, and monitored (manual or automated recording) area in accordance with the labeled storage conditions with access limited to the investigator and authorized site staff. At a minimum, daily minimum and maximum temperatures for all site storage locations must be documented and available upon request. Data for nonworking days must indicate the minimum and maximum temperatures since previously documented for all site storage locations upon return to business.
- Any excursions from the study intervention label storage conditions should be reported to Pfizer upon discovery along with any actions taken. The site should actively pursue options for returning the study intervention to the storage conditions described in the labeling, as soon as possible. Once an excursion is identified, the study intervention must be quarantined and not used until Pfizer provides permission to use the study intervention. Specific details regarding the definition of an excursion and information the site should report for each excursion will be provided to the site in the IPM.

- Any storage conditions stated in the SRSD will be superseded by the storage conditions stated on the label.
- Study interventions should be stored in their original containers.
- See the IPM for storage conditions of the study intervention once reconstituted.
- The investigator, institution, or the head of the medical institution (where applicable) is responsible for study intervention accountability, reconciliation, and record maintenance (ie, receipt, reconciliation, and final disposition records), such as the IPAL or sponsor-approved equivalent. All study interventions will be accounted for using a study intervention accountability form/record.
- Further guidance and information for the final disposition of unused study interventions are provided in the IPM. All destruction must be adequately documented. If destruction is authorized to take place at the investigator site, the investigator must ensure that the materials are destroyed in compliance with applicable environmental regulations, institutional policy, and any special instructions provided by Pfizer.

Upon identification of a product complaint, notify the sponsor within 1 business day of discovery as described in the IPM.

## 6.4.1. Preparation and Dispensing

See the IPM for instructions on how to prepare the study intervention for administration. Study intervention should be prepared and dispensed by an appropriately medically qualified and experienced member of the study staff (eg, physician, nurse, physician's assistant, nurse practitioner, pharmacy assistant/technician, or pharmacist) as allowed by local, state, and institutional guidance. A second staff member will verify the preparation and dispensing.

#### 6.5. Measures to Minimize Bias: Randomization and Blinding

#### 6.5.1. Randomization to Study Intervention

Randomization of participants to vaccine groups will proceed through the use of an IRT system. The site personnel (study coordinator or specified designee) will be required to enter or select information including but not limited to the user's ID and password, the protocol number, and the participant number. The site personnel will then be provided with a vaccine assignment, randomization number, and DU or container number when study intervention is being supplied via the IRT system. The IRT system will provide a confirmation report containing the participant number, randomization number, and DU or container number assigned. The confirmation report must be stored in the site's files.

The study-specific IRT reference manual and IPM will provide the contact information and further details on the use of the IRT system.

## **6.5.2. Blinding Arrangements**

This study is double-blinded.

## 6.5.2.1. Blinding of Study Site Personnel

The participant, study coordinator, and all site staff will be blinded.

Please refer to the IPM for further details.

## 6.5.2.2. Blinding of the Sponsor

The majority of sponsor staff will be blinded to study intervention allocation. All laboratory testing personnel performing serological assays or diagnostic assays will remain blinded to the study intervention assigned/received throughout the study.

## 6.5.3. Breaking the Blind

The IRT will be programmed with blind-breaking instructions. In case of an emergency, the investigator has the sole responsibility for determining if unblinding of a participant's vaccine assignment is warranted. Participant safety must always be the first consideration in making such a determination. If the investigator decides that unblinding is warranted, the investigator should make every effort to contact the sponsor prior to unblinding a participant's vaccine assignment unless this could delay further management of the participant. If a participant's vaccine assignment is unblinded, the sponsor must be notified within 24 hours after breaking the blind. The date and reason that the blind was broken must be recorded in the source documentation and CRF.

The study-specific IRT reference manual and IPM will provide the contact information and further details on the use of the IRT system.

#### 6.6. Study Intervention Compliance

Participants will receive study intervention directly from the investigator or designee, under medical supervision. The date and time of administration will be recorded in the source documents and in the CRF. The study intervention identification details and study participant identification will be checked and confirmed at the time of and prior to administration by a second member of the study site staff who is not the person administering the vaccine.

The site will complete the required vaccine Preparation Record located in the IPM. The use of the Preparation Record is preferred, but it does not preclude the use of an existing appropriate clinical site documentation system. The existing clinical site's documentation system should capture all pertinent/required information on the preparation and administration of the dose. This may be used in place of the Preparation Record after approval from the sponsor and/or designee.

#### 6.7. Dose Modification

Not applicable.

## 6.8. Continued Access to Study Intervention After the End of the Study

No intervention will be provided to study participants at the end of their study participation.

#### 6.9. Treatment of Overdose

For this study, any dose of study intervention greater than 1 dose of study intervention within a 24-hour time period will be considered an overdose.

There is no specific treatment for an overdose.

In the event of an overdose, the investigator should:

- Contact the medical monitor within 24 hours.
- Closely monitor the participant for any AEs/SAEs.
- Document the quantity of the excess dose as well as the duration of the overdose in the CRF.
- Overdose is reportable to Pfizer Safety only when associated with an SAE.

## **6.10. Concomitant Therapy**

#### 6.10.1. Prohibited Concomitant Vaccinations and Medications

- Licensed or nonstudy investigational RSV vaccines are prohibited at any time prior to enrollment and thereafter during the course of the study.
- Investigational vaccines and investigational drugs are prohibited within 28 days prior to enrollment and at any time during the study.

#### 6.10.2. Withholding Periods for Concomitant Vaccinations and Medications

Unless considered medically necessary, the following restrictions apply to nonstudy licensed vaccines and medications as well as COVID-19 vaccines authorized for temporary or emergency use:

- Nonstudy nonlive vaccines (including licensed or authorized COVID-19 vaccines) may not be given within 14 days before or after study intervention administration.
- Nonstudy live vaccines should not be given within 28 days before or within 28 days after study intervention administration.
- Systemic corticosteroids (≥20 mg/day of prednisone or equivalent) for ≥14 days should not be given within 28 days before study intervention administration through the conclusion of study participation.

- Chronic systemic treatment with known immunosuppressant medications should not be given within 60 days before study intervention administration through the conclusion of study participation.
- Blood/plasma products or immunoglobulin should not be given within 60 days before study intervention administration through the conclusion of study participation.
- Prophylactic antipyretics and other pain medication to prevent symptoms associated with study intervention administration are not permitted.

# 6.10.3. Permitted Nonstudy Vaccines and Medications During the Study

The following restrictions apply to permitted vaccines and medications (except when they are considered medically necessary):

- Nonstudy nonlive vaccines (including licensed or authorized COVID-19 vaccines) may be given starting 14 days after the Visit 2 study intervention administration.
- Nonstudy live vaccines may only be given after study completion.
- Inhaled/nebulized, intra-articular, intrabursal, or topical (eg, skin, eyes) corticosteroids are permitted.
- Chronic corticosteroids that do not exceed a dose equivalent to 10 mg/day of prednisone are permitted for participants with COPD or asthma
- The use of antipyretics and other pain medication to treat symptoms associated with study intervention administration is permitted.
- Medication other than that listed in Section 6.10.1 and Section 6.10.2, required for treatment of preexisting stable conditions, is permitted.

#### 6.10.4. Recording Nonstudy Vaccinations and Concomitant Medications

The following concomitant medications and vaccinations will be recorded in the CRF:

- All nonstudy vaccinations including COVID-19 vaccines, received from 28 days prior to study enrollment through conclusion of study participation.
- Immunosuppressant medications, including monoclonal antibodies.
- Systemic corticosteroids, ie, oral, IM, or IV. Do not record topical, ophthalmic, otic, inhaled, intra-articular, or intrabursal corticosteroids.
- Blood/plasma products or immunoglobulin.
# 7. DISCONTINUATION OF STUDY INTERVENTION AND PARTICIPANT DISCONTINUATION/WITHDRAWAL

## 7.1. Discontinuation of Study Intervention

It may be necessary for a participant to permanently discontinue study intervention. Reasons for permanently discontinuation of study intervention include the following: AEs, participant request, investigator request, protocol deviation, no longer meeting all the inclusion criteria, or meeting 1 or more exclusion criteria.

Discontinuation of study intervention does not represent withdrawal from the study. If study intervention is discontinued, the participant will remain in the study to be evaluated for safety. Participants who remain in the study for evaluation of safety will be contacted by telephone 1 month after their last study vaccination to record AEs.

In the event of discontinuation of study intervention, it must be documented on the appropriate CRF/in the medical records whether the participant is discontinuing further receipt of study intervention or also from study procedures, posttreatment study follow-up, and/or future collection of additional information.

# 7.2. Participant Discontinuation/Withdrawal From the Study

A participant may withdraw from the study at any time at his/her own request. Reasons for discontinuation from the study include the following:

- Refused further study procedures;
- Lost to follow-up;
- Death:
- Study terminated by sponsor;
- AEs;
- Physician decision;
- Protocol deviation;
- Participant request.

The investigator or his or her designee should capture the reason for withdrawal in the CRF for all participants.

If a participant withdraws from the study, he/she may request destruction of any remaining samples taken and not tested, and the investigator must document any such requests in the site study records and notify the sponsor accordingly.

If the participant withdraws from the study and also withdraws consent (Section 7.2.1) for disclosure of future information, no further evaluations should be performed and no additional data should be collected. The sponsor may retain and continue to use any data collected before such withdrawal of consent.

When a participant withdraws from the study because of an SAE, the SAE must be recorded on the CRF and reported on the Vaccine SAE Reporting Form.

Lack of completion of all or any of the withdrawal/early termination procedures will not be viewed as protocol deviations so long as the participant's safety was preserved.

Participants who withdraw after randomization will not be replaced.

#### 7.2.1. Withdrawal of Consent

Participants who request to discontinue receipt of study intervention will remain in the study and must continue to be followed for protocol-specified follow-up procedures. The only exception to this is when a participant specifically withdraws consent for any further contact with him or her or persons previously authorized by the participant to provide this information. Participants should notify the investigator in writing of the decision to withdraw consent from future follow-up, whenever possible. The withdrawal of consent should be explained in detail in the medical records by the investigator, as to whether the withdrawal is only from further receipt of study intervention or also from study procedures and/or posttreatment study follow-up, and entered on the appropriate CRF page. In the event that vital status (whether the participant is alive or dead) is being measured, publicly available information should be used to determine vital status only as appropriately directed in accordance with local law.

## 7.3. Lost to Follow-Up

A participant will be considered lost to follow-up if he or she repeatedly fails to return for scheduled visits and is unable to be contacted by the study site.

The following actions must be taken if a participant fails to attend a required study visit:

- The site must attempt to contact the participant and reschedule the missed visit as soon as possible. Counsel the participant on the importance of maintaining the assigned visit schedule and ascertain whether the participant wishes to and/or should continue in the study.
- Before a participant is deemed lost to follow-up, the investigator or designee must make every effort to regain contact with the participant (where possible, 3 telephone calls and, if necessary, a certified letter to the participant's last known mailing address or local equivalent methods). These contact attempts should be documented in the participant's medical record.

• Should the participant continue to be unreachable, he/she will be considered to have withdrawn from the study.

#### 8. STUDY ASSESSMENTS AND PROCEDURES

The investigator (or an appropriate delegate at the investigator site) must obtain a signed and dated ICD before performing any study-specific procedures.

The date of birth will be collected to critically evaluate the immune response and safety profile by age.

Study procedures and their timing are summarized in the SoA. Protocol waivers or exemptions are not allowed.

Safety issues should be discussed with the sponsor immediately upon occurrence or awareness to determine whether the participant should continue or discontinue study intervention.

Adherence to the study design requirements, including those specified in the SoA, is essential and required for study conduct.

All screening evaluations must be completed and reviewed to confirm that potential participants meet all eligibility criteria. The investigator will maintain a screening log to record details of all participants screened and to confirm eligibility or record reasons for screening failure, as applicable.

Every effort should be made to ensure that protocol-required tests and procedures are completed as described. However, it is anticipated that from time to time there may be circumstances outside the control of the investigator that may make it unfeasible to perform the test. In these cases, the investigator must take all steps necessary to ensure the safety and well-being of the participant. When a protocol-required test cannot be performed, the investigator will document the reason for the missed test and any corrective and preventive actions that he or she has taken to ensure that required processes are adhered to as soon as possible. The study team must be informed of these incidents in a timely manner.

For samples being collected and shipped, detailed collection, processing, storage, and shipment instructions and contact information will be provided to the investigator site prior to study initiation.

#### 8.1. Efficacy and/or Immunogenicity Assessments

#### **8.1.1.** Efficacy Assessments

Efficacy assessments are not applicable to this study.

## 8.1.2. Immunogenicity Assessments

#### 8.1.2.1. Blood Collection

Blood samples (approximately 30 mL per sample) for immunogenicity assessments will be collected from all enrolled participants just prior to each study vaccination at Visit 1 and Visit 2, and at Visit 3. The total blood sampling volume for individual participants in this study is approximately 90 mL across 2 months.

Instructions for the collection and handling of blood and serum samples will be provided in the laboratory manual. The date and time of each sample will be recorded.

The immunogenicity samples must be processed and shipped as indicated in the instructions provided to the investigator site to maintain sample integrity. Any deviations from the immunogenicity sample handling procedure (eg sample collection and processing steps, interim storage, or shipping conditions), including any actions taken, must be documented, and reported to the sponsor. On a case-by-case basis, the sponsor may make a determination as to whether sample integrity has been compromised.

## 8.1.2.2. RSV Vaccine Antibody Testing

Serum samples collected at all 3 visits will be assayed for RSV A and RSV B serum NTs CCI

RSV A and RSV B serum NTs will be determined and reported as the NT.

Sample collection, processing, storage, and shipping information can be found in the laboratory manual. All assays will be performed by Pfizer and/or at a facility designated by Pfizer.

#### 8.1.2.3. SIIV Immune Response Testing

HAI titers to the influenza strains in the SIIV administered will be determined on sera collected at Visits 1 and 2 (prior to and 1 month after SIIV administration). H3N2-neutralizing antibody titers may be determined if the H3N2 strain in the SIIV fails to hemagglutinate or hemagglutinates via neuraminidase rather than hemagglutinin, which may invalidate the HAI assay for H3N2.

# 8.1.2.4. Exploratory Assays, Including Immunogenicity Assessments and Assay **Development**

Samples remaining after completion of the planned assays from blood draws may be used for additional vaccine and infectious disease-related research. Samples may also be used for assay development, standardization, qualification, and validation. This work is critical in the development, qualification, and validation of serological assays and is required by regulatory authorities for their use in the licensure of a vaccine.

## 8.1.3. Biological Samples

Blood/serum samples will be used only for scientific research. Each sample will be labeled with a code so that the laboratory personnel testing the samples will not know the participant's identity. Samples that remain after performing assays outlined in the protocol may be stored by Pfizer. Unless a time limitation is required by local regulations or ethical requirements, the samples will be stored for up to 15 years after the end of the study and then destroyed. If allowed by the ICD, stored samples may be used for additional testing to better understand the immune responses to the vaccine(s) under study in this protocol, to inform the development of other products, and/or for vaccine-related assay work supporting vaccine programs. No testing of the participant's DNA will be performed.

The participant may request that his/her samples, if still identifiable, be destroyed at any time; however, any data already collected from those samples will still be used for this research. The biological samples may be shared with other researchers as long as confidentiality is maintained, and no testing of the participant's DNA is performed.

## 8.2. Safety Assessments

Participants will be observed for 30 minutes after vaccination, and any reactions occurring during that time will be recorded as AEs.

Planned time points for all safety assessments are provided in the SoA. Unscheduled clinical laboratory measurements may be obtained at any time during the study to assess any perceived safety issues.

#### 8.2.1. Physical Examinations

If the clinical assessment indicates that a physical examination is necessary to comprehensively evaluate the participant, a physical examination will be performed.

Physical examination findings collected during the study will be considered source data and will not be required to be reported, unless otherwise noted. Any untoward physical examination findings that are identified during the active collection period and meet the definition of an AE or SAE (Section 10.2) must be reported according to the processes in Section 8.3.1 to Section 8.3.3.

#### 8.2.2. Vital Signs

The participant's body temperature will be measured prior to each vaccination.

#### 8.2.3. Electronic Diary

Participants will be required to use an e-diary, installed on a provisioned device or as an application on a personal device, and will be asked to monitor and record local reactions, systemic events, and oral temperature each evening for 7 days following each vaccination (Day 1 through Day 7, where Day 1 is the day of vaccination). The e-diary allows recording of these assessments only within a fixed time window each day, thus providing the accurate representation of the participant's experience at that time.

Data on local reactions, systemic events, and oral temperature recorded in the e-diary will be transferred electronically to the e-diary vendor, where they will be available for review by investigators, their qualified designees, and sponsor staff at all times via a secure, restricted internet-based portal. At intervals agreed to by the vendor and Pfizer, these data will be transferred electronically to Pfizer for analysis and reporting. These data do not need to be recorded by the investigator in the CRF, except the following conditions:

- If a participant withdraws because of prompted events recorded in the e-diary, the event(s) should be recorded on the AE page of the CRF, regardless of whether the investigator considers the event(s) to be clinically significant.
- The investigator or designee must obtain stop dates for any reactions ongoing on the last day that the e-diary was completed. The stop dates should be documented in the source documents and the information entered in the CRF. In the event the reaction is ongoing at the end of the study, the reaction will be marked as ongoing.

Investigators (or appropriately qualified designees) are required to review the e-diary data online at frequent intervals to evaluate participant compliance and safety. These prospectively collected occurrences of local reactions and systemic events will be graded as described in Table 2, Table 3, and Table 4.

## 8.2.3.1. Local Reactions – Reactogenicity

Assessment of local reactions applies to both Visit 1 (RSV/placebo administration, left deltoid) and Visit 2 (RSV/placebo administration, left deltoid). Local reactions at the SIIV injection site (right deltoid) will not be recorded in the e-diary.

Following both Visit 1 and Visit 2 vaccinations (on Days 1 through 7, where Day 1 is the day of each vaccination), the participants will be asked to assess redness, swelling, and pain at the LEFT deltoid injection site and to record the symptoms in the e-diary or personal device, in the evening.

Redness and swelling will be measured by the participant and recorded in measuring device units (range: 1 to 21 and >21; an entry in the e-diary of 21 will denote  $\ge$ 21) and then categorized during analysis as mild, moderate, or severe based on the grading scale in Table 2. Measuring device units can be converted to centimeters according to the following scale: 1 measuring device unit = 0.5 cm. Pain at the injection site will be assessed by the participant as absent, mild, moderate, or severe according to Table 2.

If a severe (Grade 3) local reaction is reported in the e-diary, a telephone call with the participant should be made to ascertain further details and determine whether a site visit is clinically indicated.

Only an investigator or a qualified designee is able to classify a participant's local reaction as Grade 4, after clinical evaluation of the participant or documentation from another medically qualified source (eg, emergency room or hospital record) or, in the case of pain at the injection site only, contact with the participant. If a participant experiences a Grade 4 local reaction, the investigator must immediately notify the sponsor. A Grade 4 reaction will be collected as an AE on the CRF. The event will be graded using the AE intensity grading scale (Section 10.2.3).

If a local reaction persists beyond the end of the 7-day e-diary period, the participant will be requested to report that information and/or any new AEs that develop to the investigator. The investigator will enter this additional information in the participant's source notes and CRF.

| | Mild<br>Grade 1 | Moderate<br>Grade 2 | Severe<br>Grade 3 | Grade 4ª |
|---|---|---|---|---|
| Redness | >2.0 cm to 5.0 cm<br>(5 to 10 measuring<br>device units) | >5.0 cm to 10.0 cm<br>(11 to 20 measuring<br>device units) | >10 cm<br>(>20 measuring<br>device units) | Necrosis or exfoliative dermatitis |
| Swelling | >2.0 cm to 5.0 cm<br>(5 to 10 measuring<br>device units) | >5.0 cm to 10.0 cm<br>(11 to 20 measuring<br>device units) | >10 cm<br>(>20 measuring<br>device units) | Necrosis |
| Pain (at the injection site) | Does not interfere with activity | Interferes with activity | Prevents daily activity | Emergency room visit or hospitalization for severe pain at the |

**Table 2.** Grading Scale for Local Reactions

injection site

## 8.2.3.2. Systemic Events

Following both Visit 1 and Visit 2 vaccinations (Day 1 through Day 7, where Day 1 is the day of each vaccination), participants will be asked to assess fatigue, headache, nausea, vomiting, diarrhea, muscle pain, and joint pain and to record the symptoms in the e-diary that evening. The symptoms will be assessed by the participant according to Table 3.

If a severe systemic event is reported in the e-diary, a telephone call with the participant should be made to ascertain further details and determine whether a site visit is clinically indicated.

a. Only an investigator or qualified designee is able to classify a participant's local reaction as Grade 4, after clinical evaluation of the participant or documentation from another medically qualified source (eg, emergency room or hospital record) or, in the case of pain at the injection site only, contact with the participant. Grade 4 local reactions will be collected on the AE case report form and assessed by the investigator using the AE intensity grading scale provided in Section 10.2.3.

Only an investigator or qualified designee is able to classify a participant's systemic event as Grade 4, after clinical evaluation of the participant or documentation from another medically qualified source (eg, emergency room or hospital record) or contact with the participant. If a participant experiences a Grade 4 systemic event, the investigator must immediately notify the sponsor. Grade 4 reactions will be collected as an AE on the CRF and graded using the AE intensity grading scale (Section 10.2.3).

Further, if a systemic event persists beyond the end of the 7-day e-diary period, the participant will be requested to report that information and/or any new AEs that develop to the investigator. The investigator will enter this additional information in the participant's source notes and CRF.

**Table 3.** Grading Scale for Systemic Events

| | Mild<br>Grade 1 | Moderate<br>Grade 2 | Severe<br>Grade 3 | Grade 4ª |
|---|---|---|---|---|
| Fatigue (= tiredness) | Does not interfere with activity | Some interference with activity | Prevents daily routine activity | Emergency room visit or hospitalization for severe fatigue |
| Headache | Does not interfere with activity | Some interference with activity | Prevents daily routine activity | Emergency room visit or hospitalization for severe headache |
| Vomiting | 1 to 2 times in<br>24 hours | >2 times in<br>24 hours | Requires intravenous hydration | Emergency room visit or hospitalization for severe vomiting |
| Nausea | Does not interfere with activity | Some interference with activity | Prevents daily routine activity | Emergency room visit or hospitalization for severe nausea |
| Diarrhea | 2 to 3 loose stools in<br>24 hours | 4 to 5 loose stools<br>in 24 hours | 6 or more loose<br>stools in 24 hours | Emergency room visit or hospitalization for severe diarrhea |
| Muscle pain | Does not interfere with activity | Some interference with activity | Prevents daily routine activity | Emergency room visit or hospitalization for severe muscle pain |
| Joint pain | Does not interfere with activity | Some interference with activity | Prevents daily routine activity | Emergency room visit or hospitalization for severe joint pain |

a. Only an investigator or qualified designee is able to classify a participant's systemic event as Grade 4, after clinical evaluation of the participant or documentation from another medically qualified source (eg, emergency room or hospital record) or contact with the participant. Grade 4 systemic reactions will be collected on the AE case report form and assessed by the investigator using the AE intensity grading scale as detailed in Section 10.2.3.

## 8.2.3.3. Fever Monitoring

A digital thermometer will be given to the participant with instructions on how to measure oral temperature at home. Temperature will be collected in the evening for 7 days following each vaccination (Day 1 through Day 7, where Day 1 is the day of each vaccination) and at any time during the 7 days following vaccination that fever is suspected.

Fever is defined as an oral temperature of  $\geq 38.0^{\circ}$ C ( $\geq 100.4^{\circ}$ F). The highest temperature for each day will be recorded in the e-diary, where possible. Temperatures recorded in degrees Fahrenheit will be programmatically converted to degrees Celsius and then categorized according to the ranges shown in Table 4 during analysis.

In the event of a fever on the last day the diary was completed, temperature will be measured daily until fever has resolved (1 day of temperature <38.0°C [<100.4°F]) in order to collect a stop date in the CRF.

If a fever of  $\geq$ 39.0°C ( $\geq$ 102.1°F) is reported in the e-diary, a telephone contact with the participant should occur to ascertain further details and determine whether a site visit is clinically indicated. Only an investigator or medically qualified person is able to confirm a participant's fever as >40.0°C (>104.0°F). If a participant experiences a confirmed fever >40.0°C (>104.0°F), the investigator must immediately notify the sponsor. Grade 4 fevers will be collected on the AE CRF and assessed by the investigator using the AE intensity grading scale as detailed in Section 10.2.3.

**Table 4.** Ranges for Fever

| | Mild<br>Grade 1 | Moderate<br>Grade 2 | Severe<br>Grade 3 | Grade 4ª |
|---|---|---|---|---|
| Fever | T | >38.4°C to 38.9°C (101.2-102.0°F) | >38.9°C to 40.0°C<br>(102.1-104.0°F) | >40.0°C<br>(>104.0°F) |

a. Only an investigator or qualified designee is able to classify a participant's fever as Grade 4, after clinical evaluation of the participant, documentation from another medically qualified source (eg, emergency room or hospital record), or contact with the participant. Grade 4 fevers will be collected on the AE case report form and assessed by the investigator using the AE intensity grading scale as detailed in Section 10.2.3.

# 8.2.4. Clinical Safety Laboratory Assessments

Clinical safety laboratory assessments will not be collected in this study.

#### 8.2.5. Pregnancy Testing

Not applicable.

## 8.3. Adverse Events, Serious Adverse Events, and Other Safety Reporting

The definitions of an AE and an SAE can be found in Appendix 2.

The definitions of device-related safety events (ADEs and SADEs) can be found in Appendix 5. Device deficiencies are covered in Section 8.3.9.

AEs may arise from symptoms or other complaints reported to the investigator by the participant (or, when appropriate, by a caregiver, surrogate, or the participant's legally authorized representative), or they may arise from clinical findings of the investigator or other healthcare providers (clinical signs, test results, etc).

The investigator and any qualified designees are responsible for detecting, documenting, and recording events that meet the definition of an AE or SAE and remain responsible to pursue and obtain adequate information both to determine the outcome and to assess whether the event meets the criteria for classification as an SAE or caused the participant to discontinue the study (Section 7).

During the active collection period as described in Section 8.3.1, each participant will be questioned about the occurrence of AEs in a nonleading manner.

In addition, the investigator may be requested by Pfizer Safety to obtain specific follow-up information in an expedited fashion.

## 8.3.1. Time Period and Frequency for Collecting AE and SAE Information

The time period for actively eliciting and collecting AEs and SAEs ("active collection period") for each participant begins from the time the participant provides informed consent, which is obtained before the participant's participation in the study (ie, before undergoing any study-related procedure and/or receiving study intervention), through to study completion (Visit 3).

Follow-up by the investigator continues throughout and after the active collection period and until the AE or SAE or its sequelae resolve or stabilize at a level acceptable to the investigator.

For participants who are screen failures, the active collection period ends when screen failure status is determined.

If the participant withdraws from the study and also withdraws consent for the collection of future information, the active collection period ends when consent is withdrawn.

If a participant permanently discontinues or temporarily discontinues <u>from the</u> study because of an AE or SAE, the AE or SAE must be recorded on the CRF and the SAE reported using the Vaccine SAE Reporting Form.

Investigators are not obligated to actively seek information on AEs or SAEs after the participant has concluded study participation. However, if the investigator learns of any SAE, including a death, at any time after a participant has completed or withdrawn early from the study, and he/she considers the event to be reasonably related to the study intervention, the investigator must promptly report the SAE to Pfizer using the Vaccine SAE Reporting Form.

## 8.3.1.1. Reporting SAEs to Pfizer Safety

All SAEs occurring in a participant during the active collection period as described in Section 8.3.1 are reported to Pfizer Safety on the Vaccine SAE Reporting Form immediately upon awareness and under no circumstance should this exceed 24 hours, as indicated in Appendix 2. The investigator will submit any updated SAE data to the sponsor within 24 hours of it being available.

## 8.3.1.2. Recording Nonserious AEs and SAEs on the CRF

All nonserious AEs and SAEs occurring in a participant during the active collection period, which begins after obtaining informed consent as described in Section 8.3.1, will be recorded on the AE section of the CRF.

The investigator is to record on the CRF all directly observed and all spontaneously reported AEs and SAEs reported by the participant.

Reporting of AEs and SAEs for participants who fail screening are subject to the CRF requirements as described in Section 5.4.

## 8.3.2. Method of Detecting AEs and SAEs

The method of recording, evaluating, and assessing causality of AEs and SAEs and the procedures for completing and transmitting SAE reports are provided in Appendix 2.

Care will be taken not to introduce bias when detecting AEs and/or SAEs. Open-ended and nonleading verbal questioning of the participant is the preferred method to inquire about AE occurrences.

## 8.3.3. Follow-Up of AEs and SAEs

After the initial AE or SAE report, the investigator is required to proactively follow each participant at subsequent visits/contacts. For each event, the investigator must pursue and obtain adequate information until resolution, stabilization, the event is otherwise explained, or the participant is lost to follow-up (as defined in Section 7.3).

In general, follow-up information will include a description of the event in sufficient detail to allow for a complete medical assessment of the case and independent determination of possible causality. Any information relevant to the event, such as concomitant medications and illnesses, must be provided. In the case of a participant death, a summary of available autopsy findings must be submitted as soon as possible to Pfizer Safety.

Further information on follow-up procedures is given in Appendix 2.

## 8.3.4. Regulatory Reporting Requirements for SAEs

Prompt notification by the investigator to the sponsor of an SAE is essential so that legal obligations and ethical responsibilities toward the safety of participants and the safety of a study intervention under clinical investigation are met.

The sponsor has a legal responsibility to notify both the local regulatory authority and other regulatory agencies about the safety of a study intervention under clinical investigation. The sponsor will comply with country-specific regulatory requirements relating to safety reporting to the regulatory authority, IRBs/ECs, and investigators.

Investigator safety reports must be prepared for SUSARs according to local regulatory requirements and sponsor policy and forwarded to investigators as necessary.

An investigator who receives SUSARs or other specific safety information (eg, summary or listing of SAEs) from the sponsor will review and then file it along with the SRSD(s) for the study and will notify the IRB/EC, if appropriate according to local requirements.

# 8.3.5. Environmental Exposure, Exposure During Pregnancy or Breastfeeding, and Occupational Exposure

Environmental exposure occurs when a person not enrolled in the study as a participant receives unplanned direct contact with or exposure to the study intervention. Such exposure may or may not lead to the occurrence of an AE or SAE. Persons at risk for environmental exposure include healthcare providers, family members, and others who may be exposed. An environmental exposure may include EDP, EDB, and occupational exposure.

Any such exposure to the study intervention under study is reportable to Pfizer Safety within 24 hours of investigator awareness.

#### **8.3.5.1.** Exposure During Pregnancy

An EDP occurs if:

- A female is found to be pregnant while being exposed or having been exposed to study intervention due to environmental exposure. Below are examples of environmental EDP:
  - A female family member or healthcare provider reports that she is pregnant after having been exposed to the study intervention by injection, ingestion, inhalation, or skin contact.
  - A male family member or healthcare provider who has been exposed to the study intervention by injection, ingestion, inhalation, or skin contact then exposes his female partner prior to or around the time of conception.

The investigator must report EDP to Pfizer Safety within 24 hours of the investigator's awareness, irrespective of whether an SAE has occurred. The initial information submitted should include the anticipated date of delivery (see below for information related to termination of pregnancy).

- If EDP occurs in a participant or participant's partner, the investigator must report this information to Pfizer Safety on the Vaccine SAE Reporting Form and an EDP Supplemental Form, regardless of whether an SAE has occurred. Details of the pregnancy will be collected after the start of study intervention and until 28 days after study intervention administration (Visit 3).
- If EDP occurs in the setting of environmental exposure, the investigator must report information to Pfizer Safety using the Vaccine SAE Reporting Form and EDP Supplemental Form. Since the exposure information does not pertain to the participant enrolled in the study, the information is not recorded on a CRF; however, a copy of the completed Vaccine SAE Reporting Form is maintained in the investigator site file.

Follow-up is conducted to obtain general information on the pregnancy and its outcome for all EDP reports with an unknown outcome. The investigator will follow the pregnancy until completion (or until pregnancy termination) and notify Pfizer Safety of the outcome as a follow-up to the initial EDP Supplemental Form. In the case of a live birth, the structural integrity of the neonate can be assessed at the time of birth. In the event of a termination, the reason(s) for termination should be specified and, if clinically possible, the structural integrity of the terminated fetus should be assessed by gross visual inspection (unless preprocedure test findings are conclusive for a congenital anomaly and the findings are reported).

Abnormal pregnancy outcomes are considered SAEs. If the outcome of the pregnancy meets the criteria for an SAE (ie, ectopic pregnancy, spontaneous abortion, intrauterine fetal demise, neonatal death, or congenital anomaly), the investigator should follow the procedures for reporting SAEs. Additional information about pregnancy outcomes that are reported to Pfizer Safety as SAEs follows:

- Spontaneous abortion including miscarriage and missed abortion.
- Neonatal deaths that occur within 1 month of birth should be reported, without regard to causality, as SAEs. In addition, infant deaths after 1 month should be reported as SAEs when the investigator assesses the infant death as related or possibly related to exposure to the study intervention.

Additional information regarding the EDP may be requested by the sponsor. Further follow-up of birth outcomes will be handled on a case-by-case basis (eg, follow-up on preterm infants to identify developmental delays). In the case of paternal exposure, the investigator will provide the participant with the Pregnant Partner Release of Information Form to deliver to his partner. The investigator must document in the source documents that the participant was given the Pregnant Partner Release of Information Form to provide to his partner.

# 8.3.5.2. Exposure During Breastfeeding

EDB occurs when:

 A female is found to be breastfeeding while being exposed or having been exposed to study intervention (ie, environmental exposure). An example of environmental EDB is a female family member or healthcare provider who reports that she is breastfeeding after having been exposed to the study intervention by injection, ingestion, inhalation, or skin contact.

The investigator must report EDB to Pfizer Safety within 24 hours of the investigator's awareness, irrespective of whether an SAE has occurred. The information must be reported using the Vaccine SAE Reporting Form. When EDB occurs in the setting of environmental exposure, the exposure information does not pertain to the participant enrolled in the study, so the information is not recorded on a CRF. However, a copy of the completed Vaccine SAE Reporting Form is maintained in the investigator site file.

An exposure during breastfeeding report is not created when a Pfizer drug specifically approved for use in breastfeeding women (eg, vitamins) is administered in accord with authorized use. However, if the infant experiences an SAE associated with such a drug, the SAE is reported together with the EDB.

## 8.3.5.3. Occupational Exposure

The investigator must report any instance of occupational exposure to Pfizer Safety within 24 hours of the investigator's awareness using the Vaccine SAE Reporting Form, regardless of whether there is an associated SAE. Since the information about the occupational exposure does not pertain to a participant enrolled in the study, the information is not recorded on a CRF; however, a copy of the completed Vaccine SAE Reporting Form must be maintained in the investigator site file.

## 8.3.6. Cardiovascular and Death Events

Not applicable.

# 8.3.7. Disease-Related Events and/or Disease-Related Outcomes Not Qualifying as AEs or SAEs

Not applicable.

#### **8.3.8.** Adverse Events of Special Interest

Not applicable.

#### 8.3.9. Medical Device Deficiencies

Medical devices are being provided for use in this study for the purposes of administering the study intervention and include a PFS and vial adapter. To fulfill regulatory reporting obligations worldwide, the investigator is responsible for the detection and documentation of events meeting the definitions of device deficiency that occur during the study with such devices.

The definition of a medical device deficiency can be found in Appendix 5.

Note: AEs and/or SAEs that are associated with a medical device deficiency will follow the same processes as other AEs or SAEs, as outlined in Section 8.3.1 through 8.3.4 and Appendix 2 of the protocol.

## 8.3.9.1. Time Period for Detecting Medical Device Deficiencies

Medical device deficiencies that result in an incident will be detected, documented, and reported during all periods of the study in which the medical device is used.

Importantly, reportable device deficiencies are not limited to problems with the device itself but also include incorrect or improper use of the device and even intentional misuse, etc.

If the investigator learns of any device deficiency at any time after a participant has been discharged from the study, and such deficiency is considered reasonably related to a medical device provided for the study, the investigator will promptly notify the sponsor.

The method of documenting medical device deficiencies is provided in Appendix 5.

#### 8.3.9.2. Follow-Up of Medical Device Deficiencies

Follow-up applies to all participants, including those who discontinue study intervention.

The investigator is responsible for ensuring that follow-up includes any supplemental investigations as indicated to elucidate the nature and/or causality of the deficiency.

New or updated information will be recorded on a follow-up form with all changes signed and dated by the investigator.

#### 8.3.9.3. Prompt Reporting of Device Deficiencies to the Sponsor

When a device deficiency occurs:

- The investigator notifies the sponsor by telephone or email within 1 business day of determining that the incident meets the protocol definition of a medical device deficiency.
- The device deficiency must be recorded on the Medical Device Complaint Form.

- If an AE (either serious or nonserious) associated with the device deficiency occurs, then the AE must be entered into the AE section of the CRF.
- If an SAE associated with the device deficiency is brought to the attention of the investigator, the investigator must immediately notify Pfizer Safety of the SAE (see Section 8.3.1.1). All relevant details related to the role of the device in the event must be included in the Vaccine SAE Reporting Form as outlined in Sections 8.3.1.1 and 8.3.1.2.

The sponsor will be the contact for the receipt of device deficiency information.

## 8.3.9.4. Regulatory Reporting Requirements for Device Deficiencies

The investigator will promptly report all device deficiencies occurring with any medical device provided for use in the study in order for the sponsor to fulfill the legal responsibility to notify appropriate regulatory authorities and other entities about certain safety information relating to medical devices being used in clinical studies.

The investigator, or responsible person according to local requirements (eg, the head of the medical institution), will comply with the applicable local regulatory requirements relating to the reporting of device deficiencies to the IRB/EC.

#### 8.3.10. Medication Errors

Medication errors may result from the administration or consumption of the study intervention by the wrong participant, or at the wrong time, or at the wrong dosage strength.

Exposures to the study intervention under study may occur in clinical trial settings, such as medication errors.

| Safety Event | Recorded on the CRF | Reported on the Vaccine SAE<br>Reporting Form to Pfizer Safety<br>Within 24 Hours of Awareness |
|---|---|---|
| Medication errors | All (regardless of whether associated with an AE) | Only if associated with an SAE |

#### Medication errors include:

- Medication errors involving participant exposure to the study intervention.
- Potential medication errors or uses outside of what is foreseen in the protocol that do or do not involve the study participant.
- The administration of expired study intervention.

- The administration of an incorrect study intervention.
- The administration of an incorrect dosage.
- The administration by an incorrect route.
- The administration of study intervention that has undergone temperature excursion from the specified storage range, unless it is determined by the sponsor that the study intervention under question is acceptable for use.

Such medication errors occurring to a study participant are to be captured on the medication error page of the CRF, which is a specific version of the AE page.

In the event of a medication dosing error, the sponsor should be notified within 24 hours.

Whether or not the medication error is accompanied by an AE, as determined by the investigator, the medication error is recorded on the medication error page of the CRF and, if applicable, any associated AE(s), serious and nonserious, are recorded on the AE page of the CRF.

Medication errors should be reported to Pfizer Safety within 24 hours on a Vaccine SAE Reporting Form **only when associated with an SAE.** 

#### 8.4. Pharmacokinetics

Pharmacokinetic parameters are not evaluated in this study.

#### 8.5. Genetics

Genetics are not evaluated in this study.

#### 8.6. Biomarkers

Biomarkers are not evaluated in this study.

## 8.7. Immunogenicity Assessments

Immunogenicity assessments are described in Section 8.1.2.

#### 8.8. Health Economics

Health economics/medical resource utilization and health economics parameters are not evaluated in this study.

## 8.9. Study Procedures

# 8.9.1. Visit 1 – Vaccination 1 (Clinic, Day 1)

Before enrollment and before any study-related procedures are performed, voluntary, written study-specific informed consent will be obtained from the participant. Each signature on the ICD must be personally dated by the signatory. The investigator or his or her designee will also sign and date the ICD. A copy of the signed and dated ICD must be given to the participant. The source data must reflect that the informed consent was obtained before participation in the study.

Study procedures should be conducted in a stepwise manner as ordered below:

- Obtain written informed consent either in electronic or hard copy format from the participant before performing any study-specific procedures.
- Assign a single participant identifier using the IRT system.
- Obtain and record the participant demography (including complete date of birth [dd-Mmm-YYYY], sex, race, racial designation, and ethnicity). The full date of birth will be collected to critically evaluate the immune response and safety profile by age.
- Obtain and record any medical history of clinical significance.
- Record current or former tobacco use.
- Perform a clinical assessment. If the clinical assessment indicates that a physical examination is necessary to comprehensively evaluate the participant, perform a physical examination and record any findings in the source documents and, if clinically significant, record on the medical history CRF.
- Measure and record prevaccination body temperature.
- Obtain details of any nonstudy vaccinations as described in Section 6.10.
- Review concomitant medication use as described in Section 6.10.
- Ensure and document that all the inclusion criteria and none of the exclusion criteria are met.
- Ensure that the participant meets none of the temporary delay criteria as described in Section 5.5. If delay criteria are met, reschedule the Visit 1 blood draw and randomization/vaccination for a later date.
- Prior to vaccination, collect a blood sample of approximately 30 mL for antibody assessment.

- Obtain the participant's randomization number and study intervention kit number using the IRT system. Refer to the IRT manual for further instructions on this process.
- Issue a measuring device to measure local reactions at the **LEFT** injection site and a thermometer for recording oral temperature.
- Explain the e-diary technologies available for this study (Section 8.2.3), and assist the participant in downloading the e-diary application onto the participant's own device or if required, issue a sponsor-provisioned e-diary.
- Work with the participant to set up the device/e-diary and provide training on daily e-diary completion. Ask the participant to complete the e-diary each evening between 4:00 PM and midnight, starting on Day 1 and completing on Day 7, where Day 1 is the day of Vaccination 1.
- Qualified site staff member(s) will administer the SIIV into the deltoid muscle of the **RIGHT** arm and the study intervention into the deltoid muscle of the **LEFT** arm.
- Observe the participant for any acute reactions for at least 30 minutes after study intervention administration. Record any acute reactions, including the time of onset, in the participant's source documents, on the AE page of the CRF, and on the Vaccine SAE Reporting Form if applicable.
- Discuss contraceptive use where applicable and as described in Section 10.3.4.
- Provide participant with an ECC and instruct the participant on its use.
- Ask the participant to contact the site staff or investigator immediately if he/she experiences any of the following reactions from Day 1 to Day 7 after Vaccination 1 (where Day 1 is the day of Vaccination 1) to determine if an unscheduled reactogenicity visit is required (Section 8.9.4).
- Fever  $\ge 39.0^{\circ}\text{C} (\ge 102.1^{\circ}\text{F}).$
- Redness or swelling at the **LEFT** injection site measuring >20 measuring device units (greater than 10 cm).
- Severe pain at the **LEFT** injection site.
- Any severe systemic event.
- Any emergency room attendance or hospitalization.
- Advise the participant that study staff may make contact to obtain additional information on events entered in the e-diary.

- Advise the participant to inform the study staff of any AEs and SAEs that occur for the duration of the study as described in Section 8.3.1.
- Request that the participant bring the completed e-diary to the next visit.
- Schedule an appointment for the participant to return for the next study visit.
- Complete the source documents.
- The investigator or an authorized designee completes the CRFs and the dispenser/administrator completes the study intervention accountability records.
- Following vaccination, the investigator or appropriately qualified designee reviews the daily e-diary data online to evaluate participant compliance and as part of the ongoing safety review.

## 8.9.2. Visit 2 – Vaccination 2 (Clinic, 28 to 35 Days After Visit 1)

- Record details of any nonstudy vaccinations and concomitant medications as described in Section 6.10.4.
- Record AEs and SAEs as described in Section 8.3.1 Obtain and record any missing AE stop dates.
- Review the participant's e-diary data. Collect stop dates of any ediary events ongoing on the last day that the e-diary was completed and record stop dates in the CRF.
- Obtain the participant's body temperature.
- Ensure that none of the temporary delay criteria are met (see Section 5.5).
- Prior to Vaccination 2, collect a blood sample of approximately 30 mL for antibody assessment.
- Qualified site staff member(s) will administer a single dose of study intervention into the deltoid muscle of the LEFT arm.
- Observe the participant for any acute reactions for at least 30 minutes after study intervention administration. Record any acute reactions, including the time of onset, in the participant's source documents, on the AE page of the CRF, and on the Vaccine SAE Reporting Form if applicable.
- Discuss contraceptive use (where applicable) and as described in Section 10.3.4.

- Confirm that the e-diary is set up for Vaccination 2 and review instructions, if necessary. Ask the participant to complete the e-diary from Day 1 to Day 7, with Day 1 being the day of Vaccination 2. Provide thermometer, measuring device, or ECC, if needed.
- Ask the participant to contact the site staff or investigator immediately if he/she experiences any of the following reactions from Day 1 to Day 7 to determine if an unscheduled reactogenicity visit is required (Section 8.9.4)
- Fever  $\ge 39.0^{\circ}\text{C} (\ge 102.1^{\circ}\text{F})$ .
- Redness or swelling at the **LEFT** injection site measuring >20 measuring device units (greater than 10 cm).
- Severe pain at the **LEFT** injection site.
- Any severe systemic event.
- Any emergency room attendance or hospitalization
- Advise the participant that study staff may make contact to obtain additional information on events entered in the e-diary.
- Advise the participant to inform the study staff of any AEs and SAEs that occur for the duration of the study as described in Section 8.3.1.
- Request that the participant brings the completed e-diary to the next visit.
- Schedule an appointment for the participant to return for the final study visit.
- Complete the source documents.
- The investigator or an authorized designee completes the CRFs and the dispenser/administrator completes the study intervention accountability records.
- Following vaccination, the investigator or appropriately qualified designee reviews the daily e-diary data online to evaluate participant compliance and as part of the ongoing safety review.

## 8.9.3. Visit 3 Follow-Up After Vaccination 2 (Clinic, 28 to 35 Days After Visit 2)

- Obtain details of any nonstudy vaccinations as described in Section 6.10.
- Review concomitant medication use as described in Section 6.10.
- Collect a blood sample of approximately 30 mL for antibody assessment.

- Review the participant's e-diary data. Collect stop dates of any ediary events ongoing on the last day that the e-diary was completed and record stop dates in the CRF. Collect the sponsor-provisioned e-diary.
- Record AEs and SAEs as described in Section 8.3.1. Obtain and record any missing AE stop dates.
- Complete the source documents.
- The investigator or an authorized designee completes the CRF.

# 8.9.4. Unscheduled Reactogenicity Visits for a Grade 3 or Suspected Grade 4 Reaction

If a severe local reaction (Section 8.2.3.1), severe systemic event (Section 8.2.3.2), or fever ≥39.0°C (≥102.1°F) (Section 8.2.3.3) is reported in the e-diary, a telephone contact with the participant should occur to ascertain further details and determine whether a site visit is clinically indicated. If a suspected Grade 4 local reaction, systemic event, or fever is reported in the reactogenicity e-diary, a telephone contact or site visit should occur to confirm whether the event meets the criteria for Grade 4.

A site visit or referral to a healthcare facility should be scheduled as soon as possible to assess the extent of the reaction, unless:

- The participant is unable to attend the unscheduled visit, or
- The reaction is no longer present at the time of the contact, or
- The participant recorded an incorrect value in the e-diary (confirmation of an e-diary data entry error), or
- The investigator or appropriate designee determines that an unscheduled visit is not required.

This contact will be recorded in the participant's source notes and in the CRF.

If the participant is unable to attend the unscheduled visit, or the principal investigator or authorized designee determined it was not needed, any ongoing local reactions/systemic events must be assessed at the next study visit.

The reactogenicity events should be assessed by the investigator or a medically qualified member of the site staff, such as a study physician or a study nurse, as applicable to the investigator's local practice or healthcare facility, who will:

- Measure body temperature and record any fever (Table 4).
- If present, measure the minimum and maximum diameters of redness at the **LEFT** injection site.

- If present, measure the minimum and maximum diameters of swelling at the **LEFT** injection site.
- Assess any **LEFT** injection site pain in accordance with the reactogenicity grading scale provided in Table 2.
- Assess any systemic events (fatigue, headache, nausea, vomiting, diarrhea, muscle pain, or joint pain) that are present in accordance with the reactogenicity grading scale provided in Table 3.
- Assess for other findings associated with the reaction and record on the AE CRF, if appropriate.
- Record AEs and SAEs as described in Section 8.3.1.
- Complete the participant's source documents.
- The investigator or an authorized designee completes the unscheduled visit assessment CRF.

#### 9. STATISTICAL CONSIDERATIONS

Methodology for summary and statistical analyses of the data collected in this study is described here and further detailed in the SAP, which will be maintained by the sponsor. The SAP may modify what is outlined in the protocol where appropriate; however, any major modifications of the primary endpoint definitions or their analyses will also be reflected in a protocol amendment.

## 9.1. Statistical Hypotheses

#### 9.1.1. Estimands

The estimands corresponding to each primary, secondary, and exploratory objectives are described in Section 3.

The estimands to evaluate the immunogenicity objectives are based on the evaluable immunogenicity population (Section 9.2). These estimands estimate the vaccine effect in the hypothetical settings where participants follow the study schedules and protocol requirements as directed. Missing immunogenicity results will not be imputed, as MCAR is assumed.

In the primary safety objective evaluations, completely missing reactogenicity e-diary data will not be imputed. Missing AE dates will be imputed according to Pfizer safety rules. No other missing information will be imputed in the safety analysis.

## 9.1.2. Statistical Hypotheses

# 9.1.2.1. Statistical Hypothesis for Primary RSV Immunogenicity

The primary immunogenicity objective on immune response elicited by RSVpreF will be evaluated by the following hypothesis for both RSV A and RSV B as measured by NT:

$$H_{01}$$
:  $ln(\mu_1) - ln(\mu_2) \le ln(0.667)$ 

where ln(0.667) corresponds to a 1.5-fold margin for noninferiority and  $ln(\mu_1)$  and  $ln(\mu_2)$  are the natural log of the geometric mean of NT at 1 month after vaccination with RSVpreF for the coadministration group (Visit 2) and the sequential-administration group (Visit 3), respectively. Noninferiority will be declared if the lower limit of the 2-sided 95% CI for the GMR (coadministration group to sequential-administration group) is >0.667 for both RSV A and RSV B NTs.

## 9.1.2.2. Statistical Hypothesis for SIIV Immunogenicity

The primary immunogenicity objective on immune response elicited by SIIV will be evaluated by the following hypothesis for each strain included in SIIV:

$$H_{02}$$
:  $ln(\mu_1) - ln(\mu_2) \le ln(0.667)$ 

where ln(0.667) corresponds to a 1.5-fold margin for noninferiority, and  $ln(\mu 1)$  and  $ln(\mu 2)$  are the natural log of the geometric mean of the strain-specific HAI titers (or H3N2-neutralizing antibody titers if interpretable H3N2-HAI titers cannot be obtained) 1 month after vaccination with SIIV for the coadministration group and the sequential-administration group, respectively. Noninferiority will be declared for an influenza strain if the lower limit of the 2-sided 95% CI for the GMR (coadministration group to sequential-administration group) is >0.667. The primary SIIV immunogenicity objective of the study will be achieved if the noninferiority is met for each of the 4 influenza strains.

## 9.1.3. Multiplicity Adjustment

No multiplicity adjustment will be applied for this study. The primary objectives of noninferiority will be achieved only if the 1.5-fold equivalence criterion is met for each strain included in SIIV and for both RSV A and RSV B antigens simultaneously. Each of the 6 statistical tests (4 from the SIIV objective and 2 from the RSV objective) will use a 2-sided alpha level of 0.05.

## 9.2. Analysis Sets

Table 5. Analysis Sets

| Analysis Set | Description |
|---|---|
| Population analysis set | |
| Enrolled | All participants who have a signed ICD. |
| Randomized population | All participants who are assigned a randomization number in the IRT system. |
| Safety population | All enrolled participants who receive the study intervention. |
| Defined analysis sets | |
| Evaluable RSV immunogenicity population | <ul> <li>All participants who meet the following criteria:</li> <li>Are eligible for the study;</li> <li>Received the study interventions to which they were randomized at both Visit 1 and Visit 2;</li> <li>Had the 1-month postvaccination blood collection within an appropriate window (Visit 2 for the coadministration group and Visit 3 for the sequential-administration group);</li> <li>Had no major protocol violations from randomization through the 1-month postvaccination blood draw;</li> <li>Had at least 1 valid and determinate assay result 1 month after vaccination.</li> </ul> |
| Evaluable SIIV immunogenicity population | <ul> <li>All participants who meet the following criteria:</li> <li>Are eligible for the study;</li> <li>Received the study interventions to which they were randomized in addition to SIIV at Visit 1;</li> <li>Had the 1-month postvaccination blood collection within an appropriate window (Visit 2);</li> <li>Had no major protocol violations from randomization through the 1-month postvaccination blood draw;</li> <li>Had at least 1 valid and determinate assay result 1 month after vaccination.</li> </ul> |
| mITT immunogenicity population | All participants who were randomized and had at least 1 valid and determinate assay result at any time point after receiving study intervention. |

## 9.3. Statistical Analyses

The SAP will be developed and finalized before any analyses are performed and will describe the analyses and procedures for accounting for missing, unused, and spurious data. This section is a summary of the planned statistical analyses of the primary and secondary endpoints.

## 9.3.1. General Considerations

CIs for all endpoints in the statistical analysis will be presented as 2-sided at the 95% level unless specified otherwise.

For all the immunogenicity endpoints, the analysis will be based on the evaluable immunogenicity populations. An additional analysis will be performed based on the mITT population if there is a large enough difference in sample size between the mITT population and the evaluable immunogenicity population(s). Participants will be summarized according to the group (coadministration group and sequential-administration group) to which they were randomized.

The safety analyses will be based on the safety population. Participants will be summarized by group according to the study intervention they actually received.

# 9.3.1.1. Analyses for Binary Data

Descriptive statistics for categorical variables (eg, proportions) are the percentage (%), the numerator (n), and the denominator (N) used in the percentage calculation. The 95% CI for percentage, and for difference in percentages, may also be presented where appropriate.

The exact 95% CI for binary endpoints for each group will be computed using the F-distribution (Clopper-Pearson). 15

The 95% CI for the difference in the proportions will be computed using the Miettinen and Nurminen<sup>16</sup> method. The 95% CI will be presented in terms of percentage.

#### 9.3.1.2. Analyses for Continuous Data

Unless otherwise stated, descriptive statistics for continuous variables are n, mean, median, SD, minimum, and maximum.

#### 9.3.1.2.1. Geometric Means

Continuous immunogenicity endpoints will be logarithmically transformed for analysis. Geometric means and associated 2-sided 95% CIs will be derived by calculating group means and CIs on the natural log scale based on the t-distribution, and then exponentiating the results.

#### 9.3.1.2.2. Geometric Mean Fold Rises

GMFRs will be calculated as the group mean of the difference of logarithmically transformed assay results (later time point minus earlier time point) and exponentiating the mean. GMFRs are limited to participants with nonmissing values at both time points. The associated 2-sided 95% CIs will be obtained by constructing CIs using Student's t distribution for the mean difference on the logarithm scale and exponentiating the confidence limits.

#### 9.3.1.2.3. Geometric Mean Ratios

The GMRs will be calculated as the mean of the difference of logarithmically transformed assay results between 2 groups (coadministration group to sequential-administration group) and exponentiating the mean. Two-sided CIs will be obtained by calculating CIs using Student's t distribution for the mean difference of the logarithmically transformed assay results and exponentiating the confidence limits.

## 9.3.1.2.4. Reverse Cumulative Distribution Curves

Empirical RCDCs will plot proportions of participants with values equal to or exceeding a specified assay value versus the indicated assay value, for all observed assay values. Data points will be joined by a step function with the line first going down and then to the right to the next assay value.

# 9.3.2. Primary Endpoint(s)

Table 6. Primary Endpoint Analyses

| Endpoint | Statistical Analysis Methods |
|---|---|
| Immunogenicity | GMRs of RSV NTs in the coadministration group to the sequential-administration group for RSV A and RSV B at 1 month after vaccination with RSVpreF will be provided along with the associated 2-sided 95% CIs (Section 9.3.1.2.3). |
| | • GMRs of strain-specific HAI titers (or H3N2-neutralizing antibody titers if interpretable H3N2-HAI titers cannot be obtained) in the coadministration group to the sequential-administration group at 1 month after vaccination with SIIV will be provided along with the associated 2-sided 95% CIs (Section 9.3.1.2.3). |
| | • Using a 1.5-fold equivalence margin, equivalence will be declared if the lower bound of the 2-sided 95% CI for the GMR is greater than 0.667 for all 4 SIIV strains and for both RSV A and RSV B antigens. |
| Safety | • Descriptive statistics will be provided for each reactogenicity endpoint for RSVpreF and placebo at both vaccination visits. Local reactions (redness, swelling and pain at the injection site) and systemic events (fever, fatigue, headache, nausea, vomiting, diarrhea, muscle pain, and joint pain) from Day 1 through Day 7 after vaccination will be presented by severity and cumulatively across severity levels. Descriptive summary statistics will include counts and percentages of participants with the indicated endpoint (Section 9.3.1.1). |
| | AEs and SAEs will be categorized according to MedDRA terms. All of the AEs will be descriptively summarized by vaccine group within 1 month after each vaccination. |
| | • A 3-tier approach will be used to summarize AEs. Under this approach, AEs are classified into 1 of 3 tiers: (1) Tier 1 events are prespecified events of clinical importance and are identified in a list in the product's safety review plan; there is no Tier 1 event identified for RSVpreF at this stage; (2) Tier 2 events are those that are not Tier 1 but are considered "relatively common"; a MedDRA preferred term is defined as a Tier 2 event if there are at least 1% of participants in at least 1 vaccine group reporting the event; (3) Tier 3 events are those that are neither Tier 1 nor Tier 2 events. For both Tier 1 and Tier 2 events, the 95% CIs for the difference in the percentage of participants reporting the events between the RSVpreF group and the placebo group will be calculated using the test statistic proposed by Miettinen and Nurminen <sup>16</sup> ; in addition, for Tier 1 events, the asymptotic p-values will also be presented for the difference in the percentage of participants reporting the events, based on the same test statistic and under the assumption that the test statistic is asymptotically normally distributed. For Tier 3 events, counts and percentages for each vaccine group will be provided. |

# 9.3.3. Secondary Endpoint(s)

**Table 7.** Secondary Endpoint Analyses

| Endpoint | Statistical Analysis Methods |
|---|---|
| Immunogenicity | <ul> <li>Geometric means (at each applicable visit) and GMFRs (from before to each applicable time point after RSVpreF vaccination) of the RSV NTs and the associated 2-sided 95% CIs will be provided for each vaccine group (coadministration group vs sequential-administration group) for RSV A and RSV B (Sections 9.3.1.2.1 and 9.3.1.2.2).</li> <li>Geometric means and GMFRs of strain-specific HAI titers or H3N2-neutralizing antibody titers (if interpretable H3N2-HAI titers cannot be obtained) before vaccination and 1 month after vaccination with SIIV and the associated 2-sided 95% CIs will be summarized similarly.</li> </ul> |

# 9.3.4. Exploratory Endpoint(s)

**Table 8.** Exploratory Endpoint Analyses

| Endpoint | Statistical Analysis Methods |
|---|---|
| Immunogenicity | <ul> <li>CCI</li> <li>For each HAI strain, counts and percentages of participants with seroprotection (defined as strain-specific HAI titers ≥1:40) before vaccination and 1 month after vaccination with SIIV will be provided for each vaccine group, along with the associated Clopper-Pearson 95% CIs.</li> </ul> |
| | <ul> <li>Seroconversion is defined as an HAI titer &lt;1:10 before SIIV vaccination and an HAI titer ≥1:40 1 month after SIIV vaccination or an HAI titer ≥1:10 before vaccination and a minimum 4-fold rise in HAI titer 1 month after SIIV vaccination. For each HAI strain, counts and percentages of participants with strain-specific HAI titer seroconversion 1 month after vaccination with SIIV, along with the associated Clopper-Pearson 95% CIs, will be provided for each vaccine group.</li> <li>Seroprotection and seroconversion for NTs will be defined in the SAP, and the</li> </ul> |
| | Seroprotection and seroconversion for NTs will be defined in the SAP, and the analysis will be similar to HAI. |

## 9.4. Interim Analyses

No formal interim analysis will be conducted for this study. Only 1 analysis will be performed at the completion of the study.

# 9.5. Sample Size Determination

Table 9 presents the power to demonstrate that the immune responses induced by coadministration of RSVpreF and SIIV are noninferior to the administration of RSVpreF or SIIV alone.

For both NT and HAI assay results, it is assumed that true ratios of the coadministration group to the sequential-administration group are not larger than 0.9 (or -0.105 with the natural log scale). The SDs of the log titers are based on Study C3671001 data.

Considering this is a short study among older adults, it is reasonable to assume a 7-8% nonevaluable rate; consequently, enrolling approximately 1400 participants in the study will provide a sample size of approximately 1300 participants to be included in the evaluable population analysis. With 650 evaluable participants per vaccine group and the above assumptions, the power is 81.6% to declare noninferiority for all 4 strains included in SIIV and both RSV A and RSV B. Power was calculated with PROC POWER in SAS using the TWOSAMPLEMEANS statement.

**Table 9. Sample Size Determination** 

| Antigen | Common SD<br>(Log e Scale) <sup>a</sup> | Difference<br>(Log e Scale) | Noninferiority<br>Margin | Power to Declare<br>Noninferiority<br>(1-Sided Alpha = 0.025) |
|---|---|---|---|---|
| RSV A | 1.3 | 0.105 | 1.5-fold | 98.6% |
| RSV B | 1.4 | 0.105 | 1.5-fold | 97.1% |
| H1N1 | 1.3 | 0.105 | 1.5-fold | 98.6% |
| H3N2 | 1.7 | 0.105 | 1.5-fold | 88.9% |
| B Strain 1 | 1.3 | 0.105 | 1.5-fold | 98.6% |
| B Strain 2 | 1.3 | 0.105 | 1.5-fold | 98.6% |
| Overall power | Overall power to reject all 6 tests | | | 81.6% |

a. The reference study is C3671001. The maximum SD across all age/vaccine groups was used for each antigen/strain.

#### 10. SUPPORTING DOCUMENTATION AND OPERATIONAL CONSIDERATIONS

# 10.1. Appendix 1: Regulatory, Ethical, and Study Oversight Considerations

## 10.1.1. Regulatory and Ethical Considerations

This study will be conducted in accordance with the protocol and with the following:

- Consensus ethical principles derived from international guidelines, including the Declaration of Helsinki and CIOMS International Ethical Guidelines;
- Applicable ICH GCP guidelines;
- Applicable laws and regulations, including applicable privacy laws.

The protocol, protocol amendments, ICD, SRSD(s), and other relevant documents (eg, advertisements) must be reviewed and approved by the sponsor, submitted to an IRB/EC by the investigator, and reviewed and approved by the IRB/EC before the study is initiated.

Any amendments to the protocol will require IRB/EC approval before implementation of changes made to the study design, except for changes necessary to eliminate an immediate hazard to study participants.

Protocols and any substantial amendments to the protocol will require health authority approval prior to initiation except for changes necessary to eliminate an immediate hazard to study participants.

The investigator will be responsible for the following:

- Providing written summaries of the status of the study to the IRB/EC annually or more frequently in accordance with the requirements, policies, and procedures established by the IRB/EC;
- Notifying the IRB/EC of SAEs or other significant safety findings as required by IRB/EC procedures;
- Providing oversight of the conduct of the study at the site and adherence to requirements of 21 CFR, ICH GCP guidelines, the IRB/EC, European Regulation 536/2014 for clinical studies (if applicable), European MDR 2017/745 for clinical device research (if applicable), and all other applicable local regulations.

## 10.1.1.1. Reporting of Safety Issues and Serious Breaches of the Protocol or ICH GCP

In the event of any prohibition or restriction imposed (ie, clinical hold) by an applicable regulatory authority in any area of the world, or if the investigator is aware of any new information that might influence the evaluation of the benefits and risks of the study intervention, Pfizer should be informed immediately.

In addition, the investigator will inform Pfizer immediately of any urgent safety measures taken by the investigator to protect the study participants against any immediate hazard, and of any serious breaches of this protocol or of the ICH GCP guidelines that the investigator becomes aware of.

#### 10.1.2. Financial Disclosure

Investigators and subinvestigators will provide the sponsor with sufficient, accurate financial information as requested to allow the sponsor to submit complete and accurate financial certification or disclosure statements to the appropriate regulatory authorities. Investigators are responsible for providing information on financial interests during the study and for 1 year after completion of the study.

#### 10.1.3. Informed Consent Process

The investigator or his/her representative will explain the nature of the study, including the risks and benefits, to the participant and answer all questions regarding the study. The participant should be given sufficient time and opportunity to ask questions and to decide whether or not to participate in the trial.

Participants must be informed that their participation is voluntary. Participants will be required to sign a statement of informed consent that meets the requirements of 21 CFR 50, local regulations, ICH guidelines, privacy, and data protection requirements, where applicable, and the IRB/EC or study center.

The investigator must ensure that each study participant is fully informed about the nature and objectives of the study, the sharing of data related to the study, and possible risks associated with participation, including the risks associated with the processing of the participant's personal data.

The participant must be informed that his/her personal study-related data will be used by the sponsor in accordance with local data protection law. The level of disclosure must also be explained to the participant.

The participant must be informed that his/her medical records may be examined by Clinical Quality Assurance auditors or other authorized personnel appointed by the sponsor, by appropriate IRB/EC members, and by inspectors from regulatory authorities.

The investigator further must ensure that each study participant is fully informed about his or her right to access and correct his or her personal data and to withdraw consent for the processing of his or her personal data.

The medical record must include a statement that written informed consent was obtained before the participant was enrolled in the study and the date on which the written consent was obtained. The authorized person obtaining the informed consent must also sign the ICD.

Participants must be reconsented to the most current version of the IRB/EC-approved ICD(s) during their participation in the study as required per local regulations.

A copy of the ICD(s) must be provided to the participant.

Participants who are rescreened may be required to sign a new ICD as per IRB, local regulations, etc.

#### 10.1.4. Data Protection

All parties will comply with all applicable laws, including laws regarding the implementation of organizational and technical measures to ensure protection of participant data.

Participants' personal data will be stored at the study site in encrypted electronic and/or paper form and will be password-protected or secured in a locked room to ensure that only authorized study staff have access. The study site will implement appropriate technical and organizational measures to ensure that the personal data can be recovered in the event of disaster. In the event of a potential personal data breach, the study site will be responsible for determining whether a personal data breach has in fact occurred and, if so, providing breach notifications as required by law.

To protect the rights and freedoms of participants with regard to the processing of personal data, participants will be assigned a single, participant-specific numerical code. Any participant records or data sets that are transferred to the sponsor will contain the numerical code; participant names will not be transferred. All other identifiable data transferred to the sponsor will be identified by this single, participant-specific code. The study site will maintain a confidential list of participants who participated in the study, linking each participant's numerical code to his or her actual identity and medical record ID. In case of data transfer, the sponsor will protect the confidentiality of participants' personal data consistent with the clinical study agreement and applicable privacy laws.

#### 10.1.5. Committees Structure

#### **10.1.5.1. Data Monitoring Committee**

This study will not use a DMC.

#### 10.1.6. Dissemination of Clinical Study Data

Pfizer fulfills its commitment to publicly disclose clinical study results through posting the results of studies on www.clinicaltrials.gov (ClinicalTrials.gov), the EudraCT, and/or www.pfizer.com, and other public registries in accordance with applicable local laws/regulations. In addition, Pfizer reports study results outside of the requirements of local laws/regulations pursuant to its SOPs.

In all cases, study results are reported by Pfizer in an objective, accurate, balanced, and complete manner and are reported regardless of the outcome of the study or the country in which the study was conducted.

## www.clinicaltrials.gov

Pfizer posts clinical trial results on www.clinicaltrials.gov for Pfizer-sponsored interventional studies (conducted in patients) that evaluate the safety and/or efficacy of a product, regardless of the geographical location in which the study is conducted. These results are submitted for posting in accordance with the format and timelines set forth by US law.

#### **EudraCT**

Pfizer posts clinical trial results on EudraCT for Pfizer-sponsored interventional studies in accordance with the format and timelines set forth by EU requirements.

## www.pfizer.com

Pfizer posts public disclosure synopses (CSR synopses in which any data that could be used to identify individual participants have been removed) on www.pfizer.com for Pfizer-sponsored interventional studies at the same time the corresponding study results are posted to www.clinicaltrials.gov.

## Documents within marketing authorization packages/submissions

Pfizer complies with the EU Policy 0070, the proactive publication of clinical data to the EMA website. Clinical data, under Phase 1 of this policy, includes clinical overviews, clinical summaries, CSRs, and appendices containing the protocol and protocol amendments, sample CRFs, and statistical methods. Clinical data, under Phase 2 of this policy, includes the publishing of individual participant data. Policy 0070 applies to new marketing authorization applications submitted via the centralized procedure since 01 Jan 2015 and applications for line extensions and for new indications submitted via the centralized procedure since 01 Jul 2015.

## **Data sharing**

Pfizer provides researchers secure access to participant-level data or full CSRs for the purposes of "bona-fide scientific research" that contributes to the scientific understanding of the disease, target, or compound class. Pfizer will make data from these trials available 24 months after study completion. Participant-level data will be anonymized in accordance with applicable privacy laws and regulations. CSRs will have personally identifiable information redacted.

Data requests are considered from qualified researchers with the appropriate competencies to perform the proposed analyses. Research teams must include a biostatistician. Data will not be provided to applicants with significant conflicts of interest, including individuals requesting access for commercial/competitive or legal purposes.

## 10.1.7. Data Quality Assurance

All participant data relating to the study will be recorded on printed or electronic CRF unless transmitted to the sponsor or designee electronically (eg, laboratory data). The investigator is responsible for verifying that data entries are accurate and correct by physically or electronically signing the CRF.

Guidance on completion of CRFs will be provided in the CRF Completion Requirements document.

The investigator must ensure that the CRFs are securely stored at the study site in encrypted electronic and/or paper form and are password protected or secured in a locked room to prevent access by unauthorized third parties.

QTLs are predefined parameters that are monitored during the study. Important deviations from the QTLs and any remedial actions taken will be summarized in the clinical study report.

The investigator must permit study-related monitoring, audits, IRB/EC review, and regulatory agency inspections and provide direct access to source data documents. This verification may also occur after study completion. It is important that the investigator(s) and their relevant personnel are available during the monitoring visits and possible audits or inspections and that sufficient time is devoted to the process.

Monitoring details describing strategy, including definition of study-critical data items and processes (eg, risk-based initiatives in operations and quality such as risk management and mitigation strategies and analytical risk-based monitoring), methods, responsibilities, and requirements, including handling of noncompliance issues and monitoring techniques (central, virtual, or on-site monitoring), are provided in the data management plan and monitoring plan maintained and utilized by the sponsor or designee.

The sponsor or designee is responsible for the data management of this study, including quality checking of the data.

Records and documents, including signed ICDs, pertaining to the conduct of this study must be retained by the investigator for 15 years after study completion unless local regulations or institutional policies require a longer retention period. No records may be destroyed during the retention period without the written approval of the sponsor. No records may be transferred to another location or party without written notification to the sponsor. The investigator must ensure that the records continue to be stored securely for as long as they are maintained.

When participant data are to be deleted, the investigator will ensure that all copies of such data are promptly and irrevocably deleted from all systems.

The investigator(s) will notify the sponsor or its agents immediately of any regulatory retain notification in relation to the study. Furthermore, the investigator will cooperate with the sponsor or its agents to prepare the investigator site for the inspection and will allow the sponsor or its agent, whenever feasible, to be present during the inspection. The investigator site and investigator will promptly resolve any discrepancies that are identified between the study data and the participant's medical records. The investigator will promptly provide copies of the inspection findings to the sponsor or its agent. Before response submission to the regulatory authorities, the investigator will provide the sponsor or its agents with an opportunity to review and comment on responses to any such findings.

#### 10.1.8. Source Documents

Source documents provide evidence for the existence of the participant and substantiate the integrity of the data collected. Source documents are filed at the investigator site.

Data reported on the CRF or entered in the eCRF that are from source documents must be consistent with the source documents or the discrepancies must be explained. The investigator may need to request previous medical records or transfer records, depending on the study. Also, current medical records must be available.

Definition of what constitutes source data and its origin can be found in the monitoring plan, which is maintained by the sponsor.

Description of the use of the computerized system is documented in the data management plan, which is maintained by the sponsor.

The investigator must maintain accurate documentation (source data) that supports the information entered in the CRF.

Study monitors will perform ongoing source data verification to confirm that data entered into the CRF by authorized site personnel are accurate, complete, and verifiable from source documents; that the safety and rights of participants are being protected; and that the study is being conducted in accordance with the currently approved protocol and any other study agreements, ICH GCP guidelines, and all applicable regulatory requirements.

#### 10.1.9. Study and Site Start and Closure

The study start date is the date on which the clinical study will be open for recruitment of participants.

The first act of recruitment is the date of the first participant's first visit and will be the study start date.

The sponsor designee reserves the right to close the study site or terminate the study at any time for any reason at the sole discretion of the sponsor. Study sites will be closed upon study completion. A study site is considered closed when all required documents and study supplies have been collected and a study-site closure visit has been performed.

The investigator may initiate study-site closure at any time upon notification to the sponsor or designee/CRO if requested to do so by the responsible IRB/EC or if such termination is required to protect the health of study participants.

Reasons for the early closure of a study site by the sponsor may include but are not limited to:

- Failure of the investigator to comply with the protocol, the requirements of the IRB/EC or local health authorities, the sponsor's procedures, or the ICH GCP guidelines.
- Inadequate recruitment of participants by the investigator.
- Discontinuation of further study intervention development.

If the study is prematurely terminated or suspended, the sponsor shall promptly inform the investigators, the ECs/IRBs, the regulatory authorities, and any CRO(s) used in the study of the reason for termination or suspension, as specified by the applicable regulatory requirements. The investigator shall promptly inform the participant and should assure appropriate participant therapy and/or follow-up.

Study termination is also provided for in the clinical study agreement. If there is any conflict between the contract and this protocol, the contract will control as to termination rights.

# 10.1.10. Publication Policy

The results of this study may be published or presented at scientific meetings by the investigator after publication of the overall study results or 1 year after the end of the study (or study termination), whichever comes first.

The investigator agrees to refer to the primary publication in any subsequent publications, such as secondary manuscripts, and submits all manuscripts or abstracts to the sponsor 30 days before submission. This allows the sponsor to protect proprietary information and to provide comments, and the investigator will, on request, remove any previously undisclosed confidential information before disclosure, except for any study- or Pfizer intervention-related information necessary for the appropriate scientific presentation or understanding of the study results.

For all publications relating to the study, the investigator will comply with recognized ethical standards concerning publications and authorship, including those established by the International Committee of Medical Journal Editors.

The sponsor will comply with the requirements for publication of the overall study results covering all investigator sites. In accordance with standard editorial and ethical practice, the sponsor will support publication of multicenter studies only in their entirety and not as individual site data. In this case, a coordinating investigator will be designated by mutual agreement.
Authorship of publications for the overall study results will be determined by mutual agreement and in line with International Committee of Medical Journal Editors authorship requirements.

If publication is addressed in the clinical study agreement, the publication policy set out in this section will not apply.

#### 10.1.11. Sponsor's Qualified Medical Personnel

The contact information for the sponsor's appropriately qualified medical personnel for the study is documented in the study contact list located in the supporting study documentation/study portal or other electronic system.

To facilitate access to appropriately qualified medical personnel for study-related medical questions or problems, participants are provided with an ECC at the time of informed consent. The ECC contains, at a minimum, (a) protocol and study intervention identifiers, (b) participant's study identification number, (c) site emergency phone number active 24 hours/day, 7 days per week, and (d) Pfizer Call Center number.

The ECC is intended to augment, not replace, the established communication pathways between the investigator, site staff, and study team. The ECC is to be used by healthcare professionals not involved in the research study only, as a means of reaching the investigator or site staff related to the care of a participant. The Pfizer Call Center number should only be used when the investigator and site staff cannot be reached. The Pfizer Call Center number is not intended for use by the participant directly; if a participant calls that number directly, he or she will be directed back to the investigator site.

## 10.2. Appendix 2: Adverse Events: Definitions and Procedures for Recording, Evaluating, Follow-Up, and Reporting

#### 10.2.1. Definition of AE

#### **AE Definition**

- An AE is any untoward medical occurrence in a patient or clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention.
- Note: An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of study intervention.

#### **Events Meeting the AE Definition**

- Any abnormal laboratory test results (hematology, clinical chemistry, or urinalysis)
  or other safety assessments (eg, ECG, radiological scans, vital sign measurements),
  including those that worsen from baseline, considered clinically significant in the
  medical and scientific judgment of the investigator. Any abnormal laboratory test
  results that meet any of the conditions below must be recorded as an AE:
  - Is associated with accompanying symptoms.
  - Requires additional diagnostic testing or medical/surgical intervention.
  - Leads to a change in study dosing (outside of any protocol-specified dose adjustments) or discontinuation from the study, significant additional concomitant drug treatment, or other therapy.
- Exacerbation of a chronic or intermittent preexisting condition, including an increase in frequency and/or intensity of the condition.
- New condition detected or diagnosed after study intervention administration, even though it may have been present before the start of the study.
- Signs, symptoms, or the clinical sequelae of a suspected drug-drug interaction.
- Signs, symptoms, or the clinical sequelae of a suspected overdose of either study intervention or a concomitant medication. Overdose per se will not be reported as an AE or SAE unless it is an intentional overdose taken with possible suicidal/self-harming intent. Such overdoses should be reported regardless of sequelae.

#### **Events NOT Meeting the AE Definition**

- Any clinically significant abnormal laboratory findings or other abnormal safety assessments that are associated with the underlying disease, unless judged by the investigator to be more severe than expected for the participant's condition.
- The disease/disorder being studied or expected progression, signs, or symptoms of the disease/disorder being studied, unless more severe than expected for the participant's condition.
- Medical or surgical procedure (eg, endoscopy, appendectomy): the condition that leads to the procedure is the AE.
- Situations in which an untoward medical occurrence did not occur (social and/or convenience admission to a hospital).
- Anticipated day-to-day fluctuations of preexisting disease(s) or condition(s) present or detected at the start of the study that do not worsen.

#### 10.2.2. Definition of an SAE

An SAE is defined as any untoward medical occurrence that, at any dose, meets one or more of the criteria listed below:

#### a. Results in death

#### b. Is life-threatening

The term "life-threatening" in the definition of "serious" refers to an event in which the participant was at risk of death at the time of the event. It does not refer to an event that hypothetically might have caused death if it were more severe.

#### c. Requires inpatient hospitalization or prolongation of existing hospitalization

In general, hospitalization signifies that the participant has been admitted (usually involving at least an overnight stay) at the hospital or emergency ward for observation and/or treatment that would not have been appropriate in the physician's office or outpatient setting. Complications that occur during hospitalization are AEs. If a complication prolongs hospitalization or fulfills any other serious criteria, the event is serious. When in doubt as to whether "hospitalization" occurred or was necessary, the AE should be considered serious.

Hospitalization for elective treatment of a preexisting condition that did not worsen from baseline is not considered an AE.

## An SAE is defined as any untoward medical occurrence that, at any dose, meets one or more of the criteria listed below:

- Results in persistent or significant disability/incapacity
- The term disability means a substantial disruption of a person's ability to conduct normal life functions.
- This definition is not intended to include experiences of relatively minor medical significance, such as uncomplicated headache, nausea, vomiting, diarrhea, influenza, and accidental trauma (eg, sprained ankle), that may interfere with or prevent everyday life functions but do not constitute a substantial disruption.

#### d. Is a congenital anomaly/birth defect

## e. Is a suspected transmission via a Pfizer product of an infectious agent, pathogenic or nonpathogenic

The event may be suspected from clinical symptoms or laboratory findings indicating an infection in a participant exposed to a Pfizer product. The terms "suspected transmission" and "transmission" are considered synonymous. These cases are considered unexpected and handled as serious expedited cases by pharmacovigilance personnel. Such cases are also considered for reporting as product defects, if appropriate.

#### f. Other situations:

- Medical or scientific judgment should be exercised by the investigator in deciding
  whether SAE reporting is appropriate in other situations, such as significant medical
  events that may jeopardize the participant or may require medical or surgical
  intervention to prevent one of the other outcomes listed in the above definition.
  These events should usually be considered serious.
- Examples of such events include invasive or malignant cancers, intensive treatment in an emergency room or at home for allergic bronchospasm, blood dyscrasias or convulsions that do not result in hospitalization, or development of drug dependency or drug abuse.

## 10.2.3. Recording/Reporting and Follow-Up of AEs and/or SAEs During the Active Collection Period

#### AE and SAE Recording/Reporting

The table below summarizes the requirements for recording AEs on the CRF and for reporting SAEs on the Vaccine SAE Reporting Form to Pfizer Safety throughout the active collection period. These requirements are delineated for 3 types of events: (1) SAEs; (2) nonserious AEs; and (3) exposure to the study intervention under study during pregnancy or breastfeeding, and occupational exposure.

It should be noted that the Vaccine SAE Reporting Form for reporting of SAE information is not the same as the AE page of the CRF. When the same data are collected, the forms must be completed in a consistent manner. AEs should be recorded using concise medical terminology and the same AE term should be used on both the CRF and the Vaccine SAE Reporting Form for reporting of SAE information.

| Safety Event | Recorded on the CRF | Reported on the Vaccine SAE<br>Reporting Form to Pfizer<br>Safety Within 24 Hours of<br>Awareness |
|---|---|---|
| SAE | All | All |
| Nonserious AE | A11 | None |
| Exposure to the study intervention under study during pregnancy or breastfeeding. | All AEs or SAEs associated with EDP or EDB. Note: Instances of EDP or EDB not associated with an AE or SAE are not captured in the CRF. | All instances of EDP are reported (whether or not there is an associated SAE).* All instances of EDB are reported (whether or not there is an associated SAE).** |
| Environmental or occupational exposure to the product under study to a non-participant (not involving EDP or EDB). | None. Exposure to a study nonparticipant is not collected on the CRF. | The exposure (whether or not there is an associated AE or SAE) must be reported.*** |

<sup>\*</sup> **EDP** (with or without an associated AE or SAE): any pregnancy information is reported to Pfizer Safety using the Vaccine SAE Reporting Form and EDP Supplemental Form; if the EDP is associated with an SAE, then the SAE is reported to Pfizer Safety using the Vaccine SAE Reporting Form.

• When an AE or SAE occurs, it is the responsibility of the investigator to review all documentation (eg, hospital progress notes, laboratory reports, and diagnostic reports) related to the event.

<sup>\*\*</sup> **EDB** is reported to Pfizer Safety using the Vaccine SAE Reporting Form, which would also include details of any SAE that might be associated with the EDB.

<sup>\*\*\*</sup> Environmental or occupational exposure: AEs or SAEs associated with occupational exposure are reported to Pfizer Safety using the Vaccine SAE Reporting Form.

- The investigator will then record all relevant AE or SAE information in the CRF.
- It is not acceptable for the investigator to send photocopies of the participant's medical records to Pfizer Safety in lieu of completion of the Vaccine SAE Reporting Form/AE or SAE CRF page.
- There may be instances when copies of medical records for certain cases are requested by Pfizer Safety. In this case, all participant identifiers, with the exception of the participant number, will be redacted on the copies of the medical records before submission to Pfizer Safety.
- The investigator will attempt to establish a diagnosis of the event based on signs, symptoms, and/or other clinical information. Whenever possible, the diagnosis (not the individual signs/symptoms) will be documented as the AE or SAE.

| Assessment of Intensity | | |
|---|---|---|
| GRADE | If required on the AE page of the CRF, the investigator will use the adjectives MILD, MODERATE, SEVERE, or LIFE-THREATENING to describe the maximum intensity of the AE. For purposes of consistency, these intensity grades are defined as follows: | |
| 1 | MILD | Does not interfere with participant's usual function. |
| 2 | MODERATE | Interferes to some extent with participant's usual function. |
| 3 | SEVERE | Interferes significantly with participant's usual function. |
| 4 | LIFE-THREATENING | Life-threatening consequences; urgent intervention indicated. |

#### **Assessment of Causality**

- The investigator is obligated to assess the relationship between study intervention and each occurrence of each AE or SAE. The investigator will use clinical judgment to determine the relationship.
- A "reasonable possibility" of a relationship conveys that there are facts, evidence, and/or arguments to suggest a causal relationship, rather than a relationship cannot be ruled out.

- Alternative causes, such as underlying disease(s), concomitant therapy, and other risk factors, as well as the temporal relationship of the event to study intervention administration, will be considered and investigated.
- The investigator will also consult the IB and/or product information, for marketed products, in his/her assessment.
- For each AE or SAE, the investigator <u>must</u> document in the medical notes that he/she has reviewed the AE or SAE and has provided an assessment of causality.
- There may be situations in which an SAE has occurred, and the investigator has minimal information to include in the initial report to the sponsor. However, it is very important that the investigator always make an assessment of causality for every event before the initial transmission of the SAE data to the sponsor.
- The investigator may change his/her opinion of causality in light of follow-up information and send an SAE follow-up report with the updated causality assessment.
- The causality assessment is one of the criteria used when determining regulatory reporting requirements.
- If the investigator does not know whether or not the study intervention caused the event, then the event will be handled as "related to study intervention" for reporting purposes, as defined by the sponsor. In addition, if the investigator determines that an SAE is associated with study procedures, the investigator must record this causal relationship in the source documents and CRF, and report such an assessment in the dedicated section of the Vaccine SAE Reporting Form and in accordance with the SAE reporting requirements.

#### Follow-Up of AEs and SAEs

- The investigator is obligated to perform or arrange for the conduct of supplemental measurements and/or evaluations, as medically indicated or as requested by the sponsor, to elucidate the nature and/or causality of the AE or SAE as fully as possible. This may include additional laboratory tests or investigations, histopathological examinations, or consultation with other healthcare providers.
- If a participant dies during participation in the study or during a recognized follow-up period, the investigator will provide Pfizer Safety with a copy of any postmortem findings, including histopathology.
- New or updated information will be recorded in the originally submitted documents.
- The investigator will submit any updated SAE data to the sponsor within 24 hours of receipt of the information.

#### 10.2.4. Reporting of SAEs

#### SAE Reporting to Pfizer Safety via an Electronic Data Collection Tool

- The primary mechanism for reporting an SAE to Pfizer Safety will be the electronic data collection tool.
- If the electronic system is unavailable, then the site will use the paper SAE data collection tool (see next section) to report the event within 24 hours.
- The site will enter the SAE data into the electronic system as soon as the data become available.
- After the study is completed at a given site, the electronic data collection tool will be taken off-line to prevent the entry of new data or changes to existing data.
- If a site receives a report of a new SAE from a study participant or receives updated data on a previously reported SAE after the electronic data collection tool has been taken off-line, then the site can report this information on a paper SAE form (see next section) or to Pfizer Safety by telephone.

#### SAE Reporting to Pfizer Safety via Vaccine SAE Reporting Form

- Facsimile transmission of the Vaccine SAE Reporting Form is the preferred method to transmit this information to Pfizer Safety.
- In circumstances when the facsimile is not working, notification by telephone is acceptable with a copy of the Vaccine SAE Reporting Form sent by overnight mail or courier service.
- Initial notification via telephone does not replace the need for the investigator to complete and sign the Vaccine SAE Reporting Form pages within the designated reporting time frames.

#### 10.3. Appendix 3: Contraceptive and Barrier Guidance

#### 10.3.1. Male Participant Reproductive Inclusion Criteria

Male participants are eligible to participate if they agree to the following requirements during the intervention period and for at least 28 days after the last dose of study intervention, which corresponds to the time needed to eliminate reproductive safety risk of the study intervention(s):

• Refrain from donating sperm.

#### PLUS either:

 Be abstinent from heterosexual intercourse with a female of childbearing potential as their preferred and usual lifestyle (abstinent on a long-term and persistent basis) and agree to remain abstinent.

OR

- Must agree to use contraception/barrier as detailed below:
  - Agree to use a male condom when having sexual intercourse with a woman of childbearing potential who is not currently pregnant.

#### 10.3.2. Female Participant Reproductive Inclusion Criteria

A female participant is eligible to participate if she is not pregnant or breastfeeding, and is not a WOCBP (see definitions below in Section 10.3.3).

#### 10.3.3. Woman of Childbearing Potential

A woman is considered fertile following menarche and until becoming postmenopausal unless permanently sterile (see below).

If fertility is unclear (eg, amenorrhea in adolescents or athletes) and a menstrual cycle cannot be confirmed before the first dose of study intervention, additional evaluation should be considered.

Women in the following categories are not considered WOCBP:

- 1. Premenopausal female with 1 of the following:
  - Documented hysterectomy;
  - Documented bilateral salpingectomy;
  - Documented bilateral oophorectomy.

For individuals with permanent infertility due to an alternate medical cause other than the above, (eg, mullerian agenesis, androgen insensitivity), investigator discretion should be applied to determining study entry.

Note: Documentation for any of the above categories can come from the site personnel's review of the participant's medical records, medical examination, or medical history interview. The method of documentation should be recorded in the participant's medical record for the study.

#### 2. Postmenopausal female:

- A postmenopausal state is defined as no menses for 12 months without an alternative medical cause. In addition:
  - A high FSH level in the postmenopausal range must be used to confirm a postmenopausal state in women under 60 years of age and not using hormonal contraception or HRT.
  - A female on HRT and whose menopausal status is in doubt will be required to use one of the nonestrogen hormonal highly effective contraception methods if they wish to continue their HRT during the study. Otherwise, they must discontinue HRT to allow confirmation of postmenopausal status before study enrollment.

#### 10.3.4. Contraception Methods

As all female participants in this study are at least 65 years of age, contraceptive use is not required for females.

Refer to Section 10.3.1 for male participants.

# 10.4. Appendix 4: Liver Safety: Suggested Actions and Follow-Up Assessments Potential Cases of Drug Induced Liver Injury

Humans exposed to a drug who show no sign of liver injury (as determined by elevations in transaminases) are termed "tolerators," while those who show transient liver injury but adapt are termed "adaptors." In some participants, transaminase elevations are a harbinger of a more serious potential outcome. These participants fail to adapt and therefore are "susceptible" to progressive and serious liver injury, commonly referred to as DILI. Participants who experience a transaminase elevation above 3 × ULN should be monitored more frequently to determine if they are "adaptors" or are "susceptible."

LFTs are not required as a routine safety monitoring procedure in this study. However, should an investigator deem it necessary to assess LFTs because a participant presents with clinical signs/symptoms, such LFT results should be managed and followed as described below.

In the majority of DILI cases, elevations in AST and/or ALT precede TBili elevations (>2 × ULN) by several days or weeks. The increase in TBili typically occurs while AST/ALT is/are still elevated above 3 × ULN (ie, AST/ALT and TBili values will be elevated within the same laboratory sample). In rare instances, by the time TBili elevations are detected, AST/ALT values might have decreased. This occurrence is still regarded as a potential DILI. Therefore, abnormal elevations in either AST OR ALT in addition to TBili that meet the criteria outlined below are considered potential DILI (assessed per Hy's law criteria) cases and should always be considered important medical events, even before all other possible causes of liver injury have been excluded.

The threshold of laboratory abnormalities for a potential DILI case depends on the participant's individual baseline values and underlying conditions. Participants who present with the following laboratory abnormalities should be evaluated further as potential DILI (Hy's law) cases to definitively determine the etiology of the abnormal laboratory values:

- Participants with AST/ALT and TBili baseline values within the normal range who subsequently present with AST OR ALT values >3 × ULN AND a TBili value >2 × ULN with no evidence of hemolysis and an alkaline phosphatase value <2 × ULN or not available.
- For participants with baseline AST **OR** ALT **OR** TBili values above the ULN, the following threshold values are used in the definition mentioned above, as needed, depending on which values are above the ULN at baseline:
  - Preexisting AST or ALT baseline values above the normal range: AST or ALT values >2 times the baseline values AND >3 × ULN; or >8 × ULN (whichever is smaller).

• Preexisting values of TBili above the normal range: TBili level increased from baseline value by an amount of at least 1 × ULN **or** if the value reaches >3 × ULN (whichever is smaller).

Rises in AST/ALT and TBili separated by more than a few weeks should be assessed individually based on clinical judgment; any case where uncertainty remains as to whether it represents a potential Hy's law case should be reviewed with the sponsor.

The participant should return to the investigator site and be evaluated as soon as possible, preferably within 48 hours from awareness of the abnormal results. This evaluation should include laboratory tests, detailed history, and physical assessment.

In addition to repeating measurements of AST and ALT and TBili for suspected Hy's law cases, additional laboratory tests should include albumin, CK, direct and indirect bilirubin, GGT, PT/INR, total bile acids, and alkaline phosphatase. Consideration should also be given to drawing a separate tube of clotted blood and an anticoagulated tube of blood for further testing, as needed, for further contemporaneous analyses at the time of the recognized initial abnormalities to determine etiology. A detailed history, including relevant information, such as review of ethanol, acetaminophen/paracetamol (either by itself or as a coformulated product in prescription or over-the-counter medications), recreational drug, or supplement (herbal) use and consumption, family history, sexual history, travel history, history of contact with a jaundiced person, surgery, blood transfusion, history of liver or allergic disease, and potential occupational exposure to chemicals, should be collected. Further testing for acute hepatitis A, B, C, D, and E infection, liver imaging (eg, biliary tract), and collection of serum samples for acetaminophen/paracetamol drug and/or protein adduct levels may be warranted.

All cases demonstrated on repeat testing as meeting the laboratory criteria of AST/ALT and TBili elevation defined above should be considered potential DILI (Hy's law) cases if no other reason for the LFT abnormalities has yet been found. Such potential DILI (Hy's law) cases are to be reported as SAEs, irrespective of availability of all the results of the investigations performed to determine etiology of the LFT abnormalities.

A potential DILI (Hy's law) case becomes a confirmed case only after all results of reasonable investigations have been received and have excluded an alternative etiology.

# 10.5. Appendix 5: AEs, ADEs, SAEs, SADEs, USADEs, and Device Deficiencies Definitions and Procedures for Recording, Evaluating, Follow-Up, and Reporting in Medical Device Studies

#### **Definitions of a Medical Device Deficiency**

The definitions and procedures detailed in this appendix are in accordance with ISO 14155 and the European MDR 2017/745 for clinical device research (if applicable).

Both the investigator and the sponsor will comply with all local reporting requirements for medical devices.

The detection and documentation procedures described in this protocol apply to all sponsor medical devices provided for use in the study (see Section 6.3 for the list of sponsor medical devices).

#### 10.5.1. Definition of AE and ADE

#### **AE and ADE Definition**

- An AE is defined in Appendix 2 (Section 10.2.1).
- An ADE is defined as an AE related to the use of an investigational medical device. This definition includes any AEs resulting from insufficient or inadequate instructions for use, deployment, implantation, installation, or operation, or any malfunction of the investigational medical device as well as any event resulting from use error or from intentional misuse of the investigational medical device.

#### 10.5.2. Definition of SAE, SADE, and USADE

#### **SAE Definition**

• An SAE is defined in Appendix 2 (Section 10.2.2).

#### **SADE Definition**

- An SADE is defined as an adverse device effect that has resulted in any of the consequences characteristic of an SAE.
- Any device deficiency that might have led to an SAE if appropriate action had not been taken, intervention had not occurred, or circumstances had been less fortunate.

#### **USADE Definition**

• A USADE is a serious adverse device effect that by its nature, incidence, severity, or outcome has not been identified in the current version of the risk analysis management file.

#### 10.5.3. Definition of Device Deficiency

#### **Device Deficiency Definition**

A device deficiency is an inadequacy of a medical device with respect to its identity, quality, durability, reliability, safety, or performance. Device deficiencies include malfunctions, use errors, and inadequate information supplied by the manufacturer.

#### 10.5.4. Recording/Reporting and Follow-Up of Medical Device Deficiencies

#### **Device Deficiency Recording**

- When a device deficiency occurs, it is the responsibility of the investigator to review all documentation (eg, hospital progress notes, laboratory reports, and diagnostic reports) related to the event.
- The investigator will then record all relevant device deficiency information in the participant's medical records, in accordance with the investigator's normal clinical practice and will also capture the required information on the Medical Device Complaint form.
- It is **not** acceptable for the investigator to send photocopies of the participant's medical records to Pfizer Safety in lieu of following the reporting process described in the Medical Device Complaint form.
- There may be instances when copies of medical records for certain cases are requested by Pfizer Safety. In this case, all participant identifiers, with the exception of the participant number, will be redacted on the copies of the medical records before submission to Pfizer Safety.
- If the investigator determines that the medical device deficiency may have injured the participant (ie, the medical device deficiency is associated with an AE or SAE), then the investigator will attempt to establish a diagnosis of the event based on signs, symptoms, and/or other clinical information. Whenever possible, the diagnosis will be documented in the participant's medical record and recorded as the AE or SAE rather than the individual signs/symptoms. Requirements for recording and reporting an AE or SAE are provided in Appendix 2 (Section 10.2.3).
- For device deficiencies, it is very important that the investigator describes any corrective or remedial actions taken to prevent recurrence of the incident.
- A remedial action is any action other than routine maintenance or servicing of a medical device where such action is necessary to prevent recurrence of a device deficiency. This includes any amendment to the device design to prevent recurrence.

#### Assessment of Causality Occurring in Conjunction With a Medical Device Deficiency

- If an AE or SAE has occurred in conjunction with a medical device deficiency, the investigator must assess the relationship between each occurrence of the AE or SAE and the medical device deficiency. The investigator will use clinical judgment to determine the relationship.
- A "reasonable possibility" of a relationship conveys that there are facts, evidence, and/or arguments to suggest a causal relationship, rather than a relationship cannot be ruled out.
- Alternative causes, such as underlying disease(s), concomitant therapy, and other risk factors, as well as the temporal relationship of the event to study intervention administration will be considered and investigated.
- The investigator will also consult the IB in his/her assessment.
- For each device deficiency, the investigator <u>must</u> document in the medical notes that he/she has reviewed the device deficiency and has provided an assessment of causality.
- There may be situations in which an SAE has occurred, and the investigator has minimal information to include in the initial report to the sponsor. However, it is very important that the investigator always make an assessment of causality for every event before the initial transmission of the SAE data to the sponsor.
- The investigator may change his/her opinion of causality in light of follow-up information and send an SAE follow-up report with the updated causality assessment.
- The causality assessment is one of the criteria used when determining regulatory reporting requirements.

#### Follow-Up of Medical Device Deficiency

- The investigator is obligated to perform or arrange for the conduct of supplemental measurements and/or evaluations, as medically indicated or as requested by the sponsor to elucidate the nature and/or causality of the device deficiency as fully as possible. This may include additional laboratory tests or investigations, histopathological examinations, or consultation with other healthcare providers.
- New or updated information regarding the nature of the device deficiency will be recorded in the originally completed Medical Device Complaint form.
- New or updated information regarding any SAE that was potentially associated with the medical device deficiency will be submitted to Pfizer Safety on the Vaccine SAE Reporting Form within 24 hours of receipt of the information, according to the requirements provided in Appendix 2, Section 10.2.

#### 10.5.5. Reporting of SAEs

Reporting of an SAE to Pfizer Safety must be performed according to the processes described in Appendix 2 (Section 10.2.4).

#### 10.5.6. Reporting of SADEs

#### **SADE Reporting to Pfizer Safety**

Note: There are additional reporting obligations for medical device deficiencies that are potentially related to SAEs (ie, a SADE) that must fulfill the legal responsibility to notify appropriate regulatory authorities and other entities about certain safety information relating to medical devices being used in clinical studies.

- Any device deficiency that is associated with an SAE must be reported to the sponsor within 24 hours after the investigator determines that the event meets the definition of a device deficiency.
- The sponsor shall review all device deficiencies and determine and document in writing whether they could have led to an SAE. These shall be reported to the regulatory authorities and IRBs/ECs as required by national regulations.

#### 10.6. Appendix 6: Alternative Measures During Public Emergencies

The alternative study measures described in this section are to be followed during public emergencies, including the COVID-19 pandemic. This appendix applies for the duration of the COVID-19 pandemic and will become effective for other public emergencies only upon written notification from Pfizer.

Use of these alternative study measures is expected to cease upon the return of business as usual (including the lifting of any quarantines and travel bans/advisories).

#### 10.6.1. Telehealth Visits

In the event that in-clinic study visits cannot be conducted, every effort should be made to follow up on the safety of study participants at scheduled visits per the schedule of activities or unscheduled visits. Telehealth visits may be used to continue to assess participant safety and collect data points. Telehealth includes the exchange of healthcare information and services via telecommunication technologies (eg, audio, video, videoconferencing software) remotely, allowing the participant and the investigator to communicate on aspects of clinical care, including medical advice, reminders, education, and safety monitoring. The following assessments must be performed during a telehealth visit:

- Review and record any AEs and SAEs since the last contact. Refer to Section 8.3.
- Obtain details of any nonstudy vaccinations and concomitant medications and treatments as described in Section 6.10.
- Confirm that the participant is adhering to the contraception method(s) required in the protocol.

Study participants must be reminded to promptly notify site staff about any change in their health status.

## 10.7. Appendix 7: Criteria for Allowing Inclusion of Participants With Chronic Stable HIV, HCV, or HBV Infection

Potential participants with chronic stable HIV, HCV, or HBV infection may be considered for inclusion if they fulfill the following respective criteria:

#### **Known HIV infection**

• Confirmed stable HIV disease defined as documented viral load <50 copies/mL and CD4 count >200 cells/mm³ within 6 months before enrollment, and on stable antiretroviral therapy for at least 6 months.

#### **Known HCV infection**

• History of chronic HCV infection with evidence of sustained virological response (defined as undetectable HCV RNA) for ≥12 weeks following HCV treatment or without evidence of HCV RNA viremia (undetectable HCV viral load).

#### **Known HBV infection**

Confirmed inactive chronic HBV infection, defined as HBsAg present for ≥6 months and the following:

- HBeAg negative, anti-HBe positive
- Serum HBV DNA <2000 IU/mL
- Persistently normal ALT and/or AST levels

In those who have had a liver biopsy performed, findings that confirm the absence of significant necroinflammation.

### 10.8. Appendix 8: Abbreviations

The following is a list of abbreviations that may be used in the protocol.

| Abbreviation | Term |
|---|---|
| ADE | adverse device effect |
| AE | adverse event |
| Al(OH) <sub>3</sub> | aluminum hydroxide |
| ALT | alanine aminotransferase |
| AST | aspartate aminotransferase |
| CFR | Code of Federal Regulations |
| CHF | congestive heart failure |
| CI | confidence interval |
| CIOMS | Council for International Organizations of Medical Sciences |
| CK | creatine kinase |
| CONSORT | Consolidated Standards of Reporting Trials |
| COPD | chronic obstructive pulmonary disease |
| COVID-19 | coronavirus disease 2019 |
| CRF | case report form |
| CRO | contract research organization |
| CSR | clinical study report |
| DILI | drug-induced liver injury |
| dLIA | direct-binding Luminex immunoassay |
| DMC | data monitoring committee |
| DNA | deoxyribonucleic acid |
| DU | dispensable unit |
| EC | ethics committee |
| ECC | emergency contact card |
| ECG | electrocardiogram |
| eCRF | electronic case report form |
| EDB | exposure during breastfeeding |
| e-diary | electronic diary |
| EDP | exposure during pregnancy |
| EMA | European Medicines Agency |
| EU | European Union |
| EudraCT | European Clinical Trials Database |
| FIH | first-in-human |

| Abbreviation | Term |
|--------------|----------------------------------------------------------|
| FI-RSV | formalin-inactivated respiratory syncytial virus vaccine |
| FSH | follicle-stimulating hormone |
| GCP | Good Clinical Practice |
| GGT | gamma-glutamyl transferase |
| GMC | geometric mean concentration |
| GMFR | geometric mean fold rise |
| GMR | geometric mean ratio |
| GMT | geometric mean titer |
| HAI | hemagglutination inhibition |
| НВе | hepatitis B e |
| HBeAg | hepatitis B e antigen |
| HBsAg | hepatitis B surface antigen |
| HBV | hepatitis B virus |
| HCV | hepatitis C virus |
| HIV | human immunodeficiency virus |
| HRT | hormone replacement therapy |
| IB | investigator's brochure |
| ICD | informed consent document |
| ICH | International Council for Harmonisation |
| ID | identification |
| CCI | |
| IM | intramuscular |
| IND | investigational new drug application |
| INR | international normalized ratio |
| IPM | investigational product manual |
| IPAL | Investigational Product Accountability Log |
| IRB | institutional review board |
| IRT | interactive response technology |
| ISO | International Organization for Standardization |
| IV | intravenous |
| LFT | liver function test |
| LRTI | lower respiratory tract illness |
| LRTI-RSV | RSV-associated lower respiratory tract illness |
| MCAR | missing completely at random |
| MDR | medical device regulation |

| Abbreviation | Term |
|---|---|
| MedDRA | Medical Dictionary for Regulatory Activities |
| mITT | modified intent-to-treat |
| N/A | not applicable |
| NT | neutralizing titer |
| PFS | prefilled syringe |
| PPE | personal protective equipment |
| PT | prothrombin time |
| QTL | quality tolerance limit |
| RCDC | reverse cumulative distribution curve |
| RNA | ribonucleic acid |
| RSV | respiratory syncytial virus |
| RSV A | respiratory syncytial virus subgroup A |
| RSV B | respiratory syncytial virus subgroup B |
| RSVpreF | respiratory syncytial virus stabilized prefusion F subunit vaccine |
| RT-PCR | reverse transcription-polymerase chain reaction |
| SADE | serious adverse device effect |
| SAE | serious adverse event |
| SAP | statistical analysis plan |
| SARS-CoV-2 | severe acute respiratory syndrome coronavirus 2 |
| SD | standard deviation |
| SIIV | seasonal inactivated influenza vaccine |
| SoA | schedule of activities |
| SOP | standard operating procedure |
| SRSD | single reference safety document |
| SUSAR | suspected unexpected serious adverse reaction |
| TBD | to be determined |
| TBili | total bilirubin |
| Th2 | T-helper type 2 |
| ULN | upper limit of normal |
| US | United States |
| USADE | unanticipated serious adverse device effect |
| WOCBP | woman/women of childbearing potential |

#### 11. REFERENCES

- Hall CB, Simőes EAF, Anderson LJ. Clinical and epidemiologic features of respiratory syncytial virus. Curr Top Microbiol Immunol. 2013;372:39-57.
- <sup>2</sup> Chadha M, Hirve S, Bancej C, et al. Human respiratory syncytial virus and influenza seasonality patterns—early findings from the WHO global respiratory syncytial virus surveillance. Influenza Other Respir Viruses. 2020;14(6):638-46.
- Baker RE, Park SW, Yang W, et al. The impact of COVID-19 nonpharmaceutical interventions on the future dynamics of endemic infections. Proc Nat Acad Sci USA. 2020;117(48):30547-53.
- Murata Y, Falsey AR. Respiratory syncytial virus infection in adults. Antivir Ther. 2007;12(4 Pt B):659-70.
- Falsey AR, Hennessey PA, Formica MA, et al. Respiratory syncytial virus infection in elderly and high-risk adults. N Engl J Med. 2005;352(17):1749-59.
- Ackerson B, Tseng HF, Sy LS, et al. Severe morbidity and mortality associated with respiratory syncytial virus versus influenza infection in hospitalized older adults. Clin Infect Dis. 2019;69(2):197-203.
- Sundaram ME, Meece JK, Sifakis F, et al. Medically attended respiratory syncytial virus infections in adults aged ≥50 years: clinical characteristics and outcomes. Clin Infect Dis. 2014;58(3):342-9.
- Belongia EA, King JP, Kieke BA, et al. Clinical features, severity, and incidence of RSV illness during 12 consecutive seasons in a community cohort of adults ≥60 years old. Open Forum Infect Dis. 2018;5(12):ofy316.
- Wyffels V, Kariburyo F, Gavart S, et al. A real-world analysis of patient characteristics and predictors of hospitalization among US Medicare beneficiaries with respiratory syncytial virus infection. Adv Ther. 2020;37(3):1203-17.
- Domachowske JB, Anderson EJ, Goldstein M. The future of respiratory syncytial virus disease prevention and treatment. Infect Dis Ther. 2021;10(Suppl 1):S47-S60.
- Centers for Disease Control and Prevention. Table 1. Influenza vaccines United States, 2020-21 influenza season. Available from: https://www.cdc.gov/flu/professionals/acip/2020-2021/acip-table.htm. Accessed: 25 Aug 2021.

- National Centre for Immunisation Research and Surveillance. ATAGI recommendation for influenza vaccine in adults aged ≥65 years. Available from: https://www.ncirs.org.au/sites/default/files/2020-12/Adjuvanted%20influenza%20vaccine%20vs%20standard%20dose%20influenza%20vaccine%20GRADE%20recommendation final.pdf. Accessed: 25 Aug 2021.
- US Food and Drug Administration. Guidance for industry: toxicity grading scale for healthy adult and adolescent volunteers enrolled in preventive vaccine clinical trials. Rockville, MD: Center for Biologics Evaluation and Research; Sep 2007.
- Fluad Quad [prescribing information]. Parkville, VIC, Aus: Seqirus Pty Ltd; 2020. Available from: https://www.ebs.tga.gov.au/ebs/picmi/picmirepository.nsf/pdf?OpenAgent&id=CP-2020-PI-02419-1&d=20210816172310101. Accessed: 25 Aug 2021
- Agresti A. Introduction: distributions and inference for categorical data. Chapter 1. In: Agresti A, ed. Categorical data analysis. 2nd ed. Hoboken, NJ: John Wiley & Sons; 2002:1-35.
- Miettinen O, Nurminen M. Comparative analysis of two rates. Stat Med. 1985;4(2): 213-26.

### **Document Approval Record**

**Document Name:** C3671006 Clinical Protocol Amendment 1, Clean Copy, 29Aug2022

**Document Title:** A PHASE 3, RANDOMIZED, DOUBLE-BLIND, PLACEBO-CONTROL

LED STUDY TO EVALUATE THE SAFETY, TOLERABILITY, AND IM MUNOGENICITY OF RESPIRATORY SYNCYTIAL VIRUS PREFUSI ON F SUBUNIT VACCINE WHEN COADMINISTERED WITH SEASO NAL INACTIVATED INFLUENZA VACCINE IN ADULTS ≥65 YEARS

OF AGE

| Signed By: | Date(GMT) | Signing Capacity |
|------------|----------------------|------------------|
| PPD | 29-Aug-2022 16:11:13 | Final Approval |
| PPD | 29-Aug-2022 17:52:24 | Final Approval |